# FINAL STUDY REPORT

Title:

Retrospective multicenter study of elderly patients with ovarian cancer treated with trabectedin and PLD according to SmPC

Study Number: GEICO 105-O

Retrospective, non-interventional (observational) study

Report Version: V1 of 14 December 2022

Sponsor: Grupo Español de Investigación en Cáncer de Ovario (GEICO)

# **Clinical Coordinating Investigator:**

Dr. María Jesús Rubio – Hospital Universitario Reina Sofía (Córdoba)

# **Funding entity:**

PharmaMar

The information contained in this document is confidential and cannot be revealed to other persons without the written authorization of the Sponsor.

# **Study Information**

| Title | Retrospective multicenter study of elderly patients with ovarian cancer treated with trabectedin and PLD according to SmPC |
|---|---|
| | dedical with tradectedin and t ED according to Sim C |
| Sponsor | Grupo Español de Investigación en Cáncer de Ovario (GEICO) |
| Version identifier of the final study report | V1 of 14 December 2022 |
| Date of last version of<br>the final study report | 14 December 2022 |
| Active substance(s) | Two drugs under observation: Trabectedin Doxorubicin hydrochloride |
| Medicinal product(s) | Two drugs under observation: Trabectedin Pegylated liposomal doxorubicin |
| Marketing authorization holder | <ul> <li>PharmaMar (Trabectedin)</li> <li>Pegylated liposomal doxorubicin (various manufacturers)</li> </ul> |
| Research question and objectives | Trabectedin in combination with pegylated liposomal doxorubicin (PLD) is indicated for platinum-sensitive relapsed ovarian cancer and is an option for those patients in whom platinum is not the best option. There are some studies with trabectedin in combination with PLD in which some patients with this profile have been included, although not exclusively. Therefore, it is of interest to study the safety and efficacy profile of this treatment in elderly patients. The general objective of the study is to describe the real-life use of trabectedin + PLD in elderly patients diagnosed with platinum-sensitive relapsed ovarian cancer treated according to the Summary of Product Characteristics (SmPC). |
| | The specific objective is to evaluate real-world data about: |
| | <ul> <li>Safety profile</li> <li>Progression-free survival (PFS)</li> <li>Overall response rate (ORR) (CR+PR) according to RECIST 1.1 criteria</li> <li>Disease control rate (DCR) (CR+PR+SD)</li> <li>Overall survival (OS)</li> <li>Trabectedin + PLD treatment information</li> <li>Previous and subsequent treatments to trabectedin + PLD</li> <li>Patient characteristics and medical history</li> </ul> |
| <b>Country of study</b> | Spain |

| Author | Patricio Ledesma |
|--------|--------------------------------------|
| | Head of Clinical Operations |
| | Sofpromed Investigación Clínica, SL |
| | CRO appointed by the Sponsor (GEICO) |

# TABLE OF CONTENTS

| 1. | Ab | stract | 6 |
|-----|-----|------------------------------------------------|----|
| 2. | Lis | t of abbreviations | 10 |
| 3. | Inv | vestigators | 11 |
| 4. | Otl | her responsible parties | 12 |
| 5. | Mi | lestones | 13 |
| 6. | Ra | tionale and background | 14 |
| 7. | Res | search questions and objectives | 16 |
| 8. | Am | nendments and updates | 17 |
| 9. | Res | search methods | 18 |
| 9 | 0.1 | Study design and setting | 18 |
| 9 | 0.2 | Subjects | 18 |
| 9 | 0.3 | Variables | 18 |
| 9 | 0.4 | Data sources and measurement | 19 |
| 9 | 0.5 | Bias | 19 |
| 9 | 0.6 | Study size | 19 |
| 9 | 0.7 | Data transformation | 19 |
| 9 | 8.0 | Statistical methods | 21 |
| | 9.8 | .1 Main summary measures | 21 |
| | 9.8 | .2 Main statistical methods | 21 |
| | 9.8 | .3 Missing values | 21 |
| | 9.8 | .4 Sensitivity analyses | 21 |
| | 9.8 | .5 Amendments to the statistical analysis plan | 21 |
| 9 | 0.9 | Quality control. | 21 |
| 10. | F | Results | 23 |
| 1 | 0.1 | Participants | 23 |
| 1 | 0.2 | Descriptive data | 23 |
| 1 | 0.3 | Outcome data | 68 |
| 1 | 0.4 | Main results | 76 |
| 1 | 0.5 | Other analyses | 76 |
| 1 | 0.6 | Adverse events/adverse reactions. | 76 |
| 11. | Ι | Discussion | 85 |
| 1 | 1.1 | Key results | 85 |

| 11. | .2 Limitations | 85 |
|-----|---------------------|----|
| 11. | .3 Interpretation | 85 |
| 11. | .4 Generalisability | 85 |
| 12. | Other information | 86 |
| 13. | Conclusion | 87 |
| 14. | References | 88 |

#### 1. Abstract

#### Title

Retrospective multicenter study of elderly patients with ovarian cancer treated with trabectedin and PLD according to SmPC

### **Keywords**

Trabectedin, pegylated liposomal doxorubicin, ovarian cancer

## Rationale and background

The median age at which ovarian cancer is diagnosed is 63 years (50-75). This is still a significant adverse factor for survival results. Seventy years can be considered the lower limit for the elderly term, since most of age-related changes occur later. Because of this, this group of patients is often not included in clinical trials and sometimes they do not receive adequate treatment. Little information is available on chemotherapy treatments in elderly patients. Data on the use of first-line chemotherapy in this population (EWOC-1) have recently been published [4].

Trabectedin in combination with PLD is indicated for platinum-sensitive relapsed ovarian cancer and is an option for those patients in whom platinum is not the best option. There are some studies with trabectedin in combination with PLD in which some patients with this profile have been included, although not exclusively. Therefore, it is of interest to study the safety and efficacy profile of this treatment in elderly patients. With this information we will be able to know its real use in routine clinical practice at the national level in Spain in this population for which not much information is available.

Safety and efficacy data (e.g., PFS, ORR, OS) will be collected retrospectively in order to draw conclusions about the combination of trabectedin + PLD, as a treatment option in this patient profile.

### Research question and objectives

Trabectedin in combination with pegylated liposomal doxorubicin (PLD) is indicated for platinumsensitive relapsed ovarian cancer and is an option for those patients in whom platinum is not the best option. There are some studies with trabectedin in combination with PLD in which some patients with this profile have been included, although not exclusively. Therefore, it is of interest to study the safety and efficacy profile of this treatment in elderly patients.

The general objective of the study is to describe the real-life use of trabectedin + PLD in elderly patients diagnosed with platinum-sensitive relapsed ovarian cancer treated according to the Summary of Product Characteristics (SmPC).

The specific objective is to evaluate real-world data about:

- Safety profile
- Progression-free survival (PFS)
- Overall response rate (ORR) (CR+PR) according to RECIST 1.1 criteria
- Disease control rate (DCR) (CR+PR+SD)
- Overall survival (OS)

- Trabectedin + PLD treatment information
- Previous and subsequent treatments to trabectedin + PLD
- Patient characteristics and medical history

## Study design and setting

The study consists of a retrospective observational, multicenter study in which the fundamental exposure factor being investigated is a drug (trabectedin and PLD). The study was developed at national level with 15 sites in Spain, during a data collection period of 5 months, including patients treated with trabectedin and PLD according to the SmPC.

The main treatment observed in this study was trabectedin in combination with PLD in elderly patients with platinum-sensitive relapsed ovarian cancer according to the SmPC. The recommended dose of trabectedin plus PLD is administered every three weeks by infusion over 3 hours at a dose of 1.1 mg/m<sup>2</sup> immediately after 30 mg/m<sup>2</sup> of PLD.

### Subjects, study size, and inclusion/exclusion criteria

The sample size was determined by all patients diagnosed with platinum-sensitive relapsed ovarian cancer treated with trabectedin and PLD between January 1st 2015 and December 31st 2019.

This retrospective clinical study was planned to include approximately 45-50 patients with the referred characteristics (no formal sample size was calculated due to the observational nature of the study).

Given that the study was a multicenter study at national level in Spain, considering a percentage of failures in the collection or analysis of the samples (missing or unevaluable data) of around 10%, a sample size of 40-45 patients with evaluable data was estimated.

The study recruited women according to the following criteria:

### Inclusion criteria:

- 1. Written informed consent must be signed by all patients participating in the study who can be interviewed in the hospital (accessible, alive patients) or absence of consent sheet must be signed by the investigator. Informed consent may not be required from inaccessible patients (dead, lost, etc.) according to ethics committee permissions and applicable law for retrospective studies in Spain.
- 2. Adult women ( $\geq$ 70 years at the time of treatment initiation with trabectedin and PLD).
- 3. Histological diagnosis of platinum-sensitive relapsed ovarian cancer (PFI  $\geq$  6 months).
- 4. Treatment started with trabectedin and PLD (at least one cycle) as standard of care between January 1st 2015 and December 31st 2019.
- 5. Patients must have received at least one cycle of trabectedin + PLD.

#### Exclusion criteria:

- 1. Patients without medical record available (lost, empty or unretrievable clinical information).
- 2. Patients who explicitly refuse to participate in the study.

#### Variables and data sources

- Safety profile: All trabectedin + PLD-related hematological and non-hematological, serious and non-serious adverse events (grade, start date, end date, action taken with trabectedin and/or PLD, outcome) will be collected. In addition, adverse event treatments will be registered in the study database.
- Progression-free survival (PFS): Defined as the time in months since first trabectedin + PLD dose date until radiological progression (or death due to any cause) according to RECIST 1.1 criteria.
- Overall response rate (ORR): Defined as the number of patients having a best overall response (BOR) of complete response (CR) or partial response (PR), divided by the total number of response-evaluable patients (according to RECIST 1.1 criteria).
- Disease control rate (DCR): Defined as the percentage of patients having a complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1 criteria.
- Overall survival (OS): Defined as the number of months since first trabectedin + PLD dose date until death due to any cause. OS will be censored at the last date the patient was known to be alive.
- Trabectedin + PLD treatment information (for both drugs): Line number in which trabectedin + PLD was given, starting dose, relative dose intensity (RDI), total dose, dose management (reductions, delays, omissions, interruptions, and their reasons), number of treatment discontinuations, reasons for discontinuations, duration of treatment, treatment status (ended or ongoing), and number of cycles.
- Previous and subsequent treatments to trabectedin + PLD: Number of previous/subsequent treatments, type, date, previous antiangiogenic agents, and clinical results of treatments before and after trabectedin + PLD.
- Patient characteristics and medical history: Sex, age, ECOG, platinum sensitivity, platinum-free interval (PFI), progression free survival (PFS), mutational status (*BRCA1*, *BRCA2*, and in other HRR genes [germline/somatic] and variant classification [pathogenic, probably pathogenic, or VOUS]), histology, tumor grade and number of previous relapses.

These data were obtained from the participating hospitals per local practice (clinical records, local reports).

#### **Results**

Between November 2021 and June 2022, 43 patients were recruited with median age 74 years (70-86). At initial diagnosis, most common FIGO stages were IIIC (51.2%), IVB (11.6%), and IIIB (7.0%). Before trabectedin+PLD (baseline), patients had ECOG performance status 0, 1, or 2 (34.1%, 41.5%, and 9.8%) and 81.4% had measurable disease. The median number of previous lines was 2 (1-6). The initial dose of trabectedin was 1.1 mg/m² in 76.7% of patients (16.3% with <1.1 and 4.7% with >1.1 mg/m²) while 76.7% of patients had PLD at 30 mg (18.6% with <30 mg and 2.3% with >30 mg). The median of trabectedin+PLD cycles was 5 (1-21) and 53.5% of patients had at least one cycle delayed. All patients ended treatment for the following reasons: patient's decision (7.0%), doctor's decision (23.3%), disease progression (39.5%), toxicity (23.83%) and 7.0% due to other factors. Median PFS for the trabectedin+PLD combination was 7.7 months (95% CI 4.4-9.4) with best overall response rates of 4 CR (9.3%), 14 PR (32.6%), 13 SD (30.2%), and 5 PD (11.6%). Median overall survival (OS) was 19.5 months (95% CI 12.8-27.2). Overall, the most common G3-4 hematological events were neutropenia (23.3%), thrombocytopenia (7.0%), and anemia (2.3%),

being asthenia (11.6%), mucositis (4.7%), and transaminitis (4.7%) the most frequent G3 non-hematological toxicities.

#### **Discussion**

The safety profile of the trabectedin+PLD combination for elderly women in real-life setting is manageable and efficacy results are comparable to those of previous clinical trials.

# **Marketing Authorization Holder**

### PharmaMar

## Names and affiliations of principal investigators

- 1. María Jesús Rubio Hospital Universitario Reina Sofía de Córdoba (Coordinating Investigator)
- 2. Blanca Hernando Fernández Hospital Universitario de Burgos
- 3. Eva Guerra Hospital Universitario Ramón y Cajal
- 4. Anna Carbó Instituto Català d'Oncologia (ICO)
- 5. Luis Miguel de Sande Hospital Universitario de León
- 6. Arancha Manzano Hospital Clínico San Carlos
- 7. Alba González-Haba Hospital Universitario de Badajoz
- 8. Alfonso Yubero-Esteban Hospital Clínico Universitario Lozano Blesa
- 9. María del Mar Gordon Hospital Universitario de Jerez de la Frontera
- 10. Diego Soto de Prado Hospital Clínico de Valladolid
- 11. Ignacio Romero Fundación Instituto Valenciano de Oncología
- 12. Purificación Estévez Hospital Universitario Virgen del Rocío
- 13. Carlos E. Robles Hospital Virgen de Valme
- 14. Jerónimo Martínez Hospital Clínico Universitario Virgen de la Arrixaca
- 15. Miguel Corbellas Hospital Universitario Dr. Peset

### 2. List of abbreviations

- AE: Adverse Event
- CM: Concomitant Medication
- CR: Complete Response
- CRO: Clinical Research Organization
- ECOG: Eastern Cooperative Oncology Group
- E-CRF: Electronic Case Report Form
- GEICO: Grupo Español de Investigación en Cáncer de Ovario
- ICF: Informed Consent Form
- KM: Kaplan-Meier
- MH: Medical History
- ORR: Overall Response Rate
- PFS: Progression-Free Survival
- PIS: Patient Information Sheet
- PR: Partial Response
- RECIST: Response Evaluation Criteria in Solid Tumors
- SD: Stable Disease

## 3. Investigators

- 1. María Jesús Rubio Hospital Universitario Reina Sofía de Córdoba (Coordinating Investigator)
- 2. Blanca Hernando Fernández Hospital Universitario de Burgos
- 3. Eva Guerra Hospital Universitario Ramón y Cajal
- 4. Anna Carbó Instituto Català d'Oncologia (ICO)
- 5. Luis Miguel de Sande Hospital Universitario de León
- 6. Arancha Manzano Hospital Clínico San Carlos
- 7. Alba González-Haba Hospital Universitario de Badajoz
- 8. Alfonso Yubero-Esteban Hospital Clínico Universitario Lozano Blesa
- 9. María del Mar Gordon Hospital Universitario de Jerez de la Frontera
- 10. Diego Soto de Prado Hospital Clínico de Valladolid
- 11. Ignacio Romero Fundación Instituto Valenciano de Oncología
- 12. Purificación Estévez Hospital Universitario Virgen del Rocío
- 13. Carlos E. Robles Hospital Virgen de Valme
- 14. Jerónimo Martínez Hospital Clínico Universitario Virgen de la Arrixaca
- 15. Miguel Corbellas Hospital Universitario Dr. Peset

# 4. Other responsible parties

The Sponsor of this study was the Grupo Español de Investigación en Cancer de Ovario (GEICO).

# 5. Milestones

| Milestone | Planned date | Actual date | Comments |
|-----------------|-----------------|------------------|---------------------|
| Start of data | 1 November 2021 | 29 November 2021 | |
| collection | | | |
| End of data | 31 March 2022 | 10 June 2022 | Includes data |
| collection | | | cleaning period. |
| | | | Delay caused by the |
| | | | need of issuing |
| | | | additional queries. |
| Final report of | 30 June 2022 | 14 December 2022 | Delay caused by the |
| study results | | | need of issuing |
| | | | additional queries. |

### 6. Rationale and background

Ovarian cancer is a devastating disease, being the fourth leading cause of cancer death in women. Its incidence increases at menopause, the mean age at diagnosis is 63 years. This is still a significant adverse factor for survival results, therefore better treatments are needed for older patients [1].

Aging is the progressive reduction of the functional reserve of multiple organ systems, as the result of spontaneous depletion and environmental influences. Seventy years of age can be considered the lower limit of senescence because most age-related changes occur after senescence.

Sabatier, Renaud, et al published a study "Prognostic factors for epithelial ovarian epithelial cancer in the elderly: a case-control study" in which they conclude that the prognosis of ovarian cancer is worse for older women, due to the fact that they are more frequently suboptimally tretated. In this study, no correlation could be observed between geriatric factors and the achievement of surgery or chemotherapy. Therefore, the treatment decision should be based on an objective geriatric evaluation to improve the outcome in this population [2].

GOG conducted an observational study (GOG 273) of chemotherapy toxicity in elderly patients with ovarian, primary peritoneal, or fallopian tube carcinoma. 290 patients were enrolled between August 2011 and Dec 2019. Patients receive chemotherapy comprising carboplatin, paclitaxel, and colony stimulating factors (regimen 1) or carboplatin alone (regimen 2) every 21 days for 4 cycles as chosen by their physicians and / or patients. Patients may undergo additional surgery and / or chemotherapy at the discretion of the treating physician. Baseline blood tests are drawn at 1, 6, and 24 hours of each cycle for pharmacokinetic studies. The quality of life of the patients is assessed using the FACT-O, FACT-Ntx, IADL questionnaires and the ability to complete the social activity questionnaires at the beginning of the study, before cycles 1 and 3, and after 3 to 6 weeks after completing treatment. Nutritional status, such as body mass index and weight loss, and comorbidity and hearing impairment are also assessed. They conclude that patients with a higher baseline IADL (instrumental activities of daily living) score (more independent) were more likely to complete 4 cycles of chemotherapy and less likely to experience grade 3 or higher toxicity [3].

The results of the EWOC-1 study, a randomized study to evaluate 3 regimens of 1st-line chemotherapy in vulnerable elderly patients diagnosed with ovarian cancer (A GCIG-ENGOT-GINECO study) have recently been published, concluding after comparing 3 chemotherapy regimens (two combinations of carboplatin + paclitaxel and the third with carboplatin alone), that monotherapy is less active and vulnerable patients have less survival than with combination regimens. Therefore, even elderly patients should be offered a carboplatin + paclitaxel regimen [4].

Currently, there are few studies that collect data on ovarian cancer in this population exclusively and in second or later lines.

In clinical trials, a part of the population affected by the disease (elderly) is not usually included. This patient profile is more common in daily clinical practice: older patients, with ECOG or PS 1-2, with comorbidities, polymedicated, etc. Around 23% of ovarian cancer patients are 70 years or older [5] and their prognosis so far tends to be worse overall, probably due to the misperception of the possibilities of optimal surgery and adequate systemic treatment.

Trabectedin in combination with pegylated liposomal doxorubicin (PLD) is indicated for the treatment of patients with recurrent platinum-sensitive ovarian cancer following the results of study OVA-301 [6]. When choosing a therapy in recurrent disease, we must not only take into account the

platinum free interval, but also the morbidities, toxicities, number of previous platinum lines, response to the last line, *BRCA* mutational status, etc. [7]. The results of the real-life European NIMES-ROC study consistently support that trabectedin + PLD is active in patients with platinum-sensitive recurrent ovarian cancer with an acceptable and manageable safety profile. The overall findings appear to be consistent with those previously observed in a randomized controlled clinical phase III trial and further support the use of trabectedin + PLD for heavily pre-treated patients with platinum-sensitive recurrent ovarian cancer [8].

In the OVA-301 study [9] and the real-life study, NIMES ROC [8], some patients with these characteristics (62-86 years) were included, so it is considered that it would be of interest to collect retrospective data from safety and efficacy at the national level to have information on the use of trabectedin in combination with PLD in daily clinical practice in elderly patients, since this is not currently available in this population.

Currently the data that are available in the population of elderly women with recurrent ovarian cancer are through non-pre-planned sub-analyzes, that is, there is no study that specifically collects the data of this profile of patients.

Oza et al. (ROSiA study) explored the efficacy and safety of bevacizumab in patients older than 70 years compared to a young population with newly diagnosed ovarian cancer. 12% of the patients included were 70 years or older, had greater comorbidities than the young population (hypertension, stage IV, ECOG greater than 1). Older patients experienced a higher incidence of adverse effects of all grades compared to the younger profile. Regarding progression-free survival at two years, the results obtained are similar between the two populations despite having a worse prognosis [10]. In the platinum-resistant elderly population, there are data from the AURELIA study subanalysis, where 37% were 65 years or older. The median PFS and response rate were similar between those <65 and ≥65 years. Grade 2 and 3 hypertension were more common in the older than 65 age group [11].

Olaparib has been studied in this population after an analysis of 8 prospective studies. Data were collected from 398 patients (78 of them aged 65 years or older), the majority had received  $\geq$  5 prior lines of chemotherapy. Tolerability and toxicity of olaparib was similar between women  $\geq$  65 years and  $\leq$  65 years of age treated for advanced recurrent ovarian cancer [12].

Regarding trabectedin, the data available are from the patients included in the phase III OVA-301 trial and in the real-life study NIMES ROC [8]. Although this population is not exclusively analyzed, patients older than 65 years and polytreated have been included [8,9]. Vergote et al., analyzed the safety profile in the population older than 65 years included in the OVA-301. There were no marked differences by age in the safety profile/tolerability of trabectedin + PLD, except for more fatigue in the older subset (≥ 65 years) compared with younger patients (< 65 years) [13]. Therefore, it would be of interest to collect data on the safety and efficacy of trabectedin in combination with PLD in elderly patients with advanced relapsed ovarian cancer to obtain information on daily clinical practice at the national level in this subgroup of patients.

## 7. Research questions and objectives

Trabectedin in combination with pegylated liposomal doxorubicin (PLD) is indicated for platinum-sensitive relapsed ovarian cancer and is an option for those patients in whom platinum is not the best option. There are some studies with trabectedin in combination with PLD in which some patients with this profile have been included, although not exclusively. Therefore, it is of interest to study the safety and efficacy profile of this treatment in elderly patients.

The general objective of the study was to describe the real-life use of trabectedin + PLD in elderly patients diagnosed with platinum-sensitive relapsed ovarian cancer treated according to the Summary of Product Characteristics (SmPC).

The specific objective was to evaluate real-world data about:

- Safety profile
- Progression-free survival (PFS)
- Overall response rate (ORR) (CR+PR) according to RECIST 1.1 criteria
- Disease control rate (DCR) (CR+PR+SD)
- Overall survival (OS)
- Trabectedin + PLD treatment information
- Previous and subsequent treatments to trabectedin + PLD
- Patient characteristics and medical history

### 8. Amendments and updates

One amendment was performed to generate protocol version 2.0 of 27 October 2021, which included the following changes:

# 5.3 Population.

- Inclusion criteria 2: ≥70 years at the time of treatment initiation with trabectedin and PLD (not the time of initial diagnosis).
- Inclusion criteria 3 has been clarified in terms of platinum sensitivity, specifying that PFI must be ≥ 6 months.
- Exclusion criteria 3: Life expectancy < 3 months has been deleted as it is not applicable for a retrospective observational study.

PFI was clarified to "Platinum Free-Interval", and PFS as "Progression Free-Survival" in all corresponding sections.

#### 9. Research methods

# 9.1 Study design and setting

The study consisted of a retrospective observational, multicenter study in which the fundamental exposure factor being investigated was a drug (trabectedin and PLD). The study was developed at national level with 15 sites in Spain, during a data collection period of 5 months, including patients treated with trabectedin and PLD according to the SmPC.

The main treatment observed in this study was trabectedin in combination with PLD in elderly patients with platinum-sensitive relapsed ovarian cancer according to the SmPC. The recommended dose of trabectedin plus PLD was administered every three weeks by infusion over 3 hours at a dose of 1.1 mg/m<sup>2</sup> immediately after 30 mg/m<sup>2</sup> of PLD.

# 9.2 Subjects

The study recruited women according to the following criteria:

### Inclusion criteria:

- 1. Written informed consent must be signed by all patients participating in the study who can be interviewed in the hospital (accessible, alive patients) or absence of consent sheet must be signed by the investigator. Informed consent may not be required from inaccessible patients (dead, lost, etc.) according to ethics committee permissions and applicable law for retrospective studies in Spain.
- 2. Adult women (≥70 years at the time of treatment initiation with trabectedin and PLD).
- 3. Histological diagnosis of platinum-sensitive relapsed ovarian cancer (PFI  $\geq$  6 months).
- 4. Treatment started with trabectedin and PLD (at least one cycle) as standard of care between January 1st 2015 and December 31st 2019.
- 5. Patients must have received at least one cycle of trabectedin + PLD.

#### Exclusion criteria:

- 1. Patients without medical record available (lost, empty or unretrievable clinical information).
- 2. Patients who explicitly refuse to participate in the study.

### 9.3 Variables

- Safety profile: All trabectedin + PLD-related hematological and non-hematological, serious and non-serious adverse events (grade, start date, end date, action taken with trabectedin and/or PLD, outcome) will be collected. In addition, adverse event treatments will be registered in the study database.
- Progression-free survival (PFS): Defined as the time in months since first trabectedin + PLD dose date until radiological progression (or death due to any cause) according to RECIST 1.1 criteria.
- Overall response rate (ORR): Defined as the number of patients having a best overall response (BOR) of complete response (CR) or partial response (PR), divided by the total number of response-evaluable patients (according to RECIST 1.1 criteria).

- Disease control rate (DCR): Defined as the percentage of patients having a complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1 criteria.
- Overall survival (OS): Defined as the number of months since first trabectedin + PLD dose date until death due to any cause. OS will be censored at the last date the patient was known to be alive.
- Trabectedin + PLD treatment information (for both drugs): Line number in which trabectedin + PLD was given, starting dose, relative dose intensity (RDI), total dose, dose management (reductions, delays, omissions, interruptions, and their reasons), number of treatment discontinuations, reasons for discontinuations, duration of treatment, treatment status (ended or ongoing), and number of cycles.
- Previous and subsequent treatments to trabectedin + PLD: Number of previous/subsequent treatments, type, date, previous antiangiogenic agents, and clinical results of treatments before and after trabectedin + PLD.
- Patient characteristics and medical history: Sex, age, ECOG, platinum sensitivity, platinum-free interval (PFI), progression free survival (PFS), mutational status (*BRCA1*, *BRCA2*, and in other HRR genes [germline/somatic] and variant classification [pathogenic, probably pathogenic, or VOUS]), histology, tumor grade and number of previous relapses.

### 9.4 Data sources and measurement

The data collected in this study included family history characteristics, clinical-pathological features of the tumor, treatment approaches (including therapies before and after the main treatment under study), safety and efficacy information, and long-term outcomes. These data were obtained from the participating hospitals per local practice (clinical records, local reports).

9.5 Bias

Since this was a retrospective observational study, no sources of bias were identified.

9.6 Study size

The sample size was determined by all patients diagnosed with platinum-sensitive relapsed ovarian cancer treated with trabectedin and PLD between January 1st 2015 and December 31st 2019.

This retrospective clinical study was planned to include approximately 45-50 patients with the referred characteristics (no formal sample size was calculated due to the observational nature of the study).

Given that the study was a multicenter study at national level in Spain, considering a percentage of failures in the collection or analysis of the samples (missing or unevaluable data) of around 10%, a sample size of 40-45 patients with evaluable data was estimated.

9.7 Data transformation

### **Stratification Factors**

No particular stratification factors were used.

### **Patients Characteristics**

The information of patients such as age, sex, race and other baseline characteristics were summarized

### **Exposure**

All data collected that was not free text was reported: mean starting dose, number of dose reductions, reasons for reductions, number of treatment discontinuations, reasons for discontinuations, and duration of treatment.

### **Concomitant Medications (CMs) and Medical History (MH)**

The CMs were presented in the summary using frequency counts and percentages. When summarizing the number and percentage of subjects with some concomitant medications, subjects with multiple occurrences of the same CM were counted only once.

In MH all data collected that was not free text was reported: number of previous relapses, number of previous chemotherapy regimens, types of treatments received (chemotherapy, targeted therapies), prior maintenance or with maintenance, treatment-free interval (platinum-based chemotherapy, non-platinum-based chemotherapy, targeted therapy).

### **Initial Ovarian Cancer Diagnosis**

The information of initial diagnosis such as age, tumor histology, and FIGO stage was summarized.

### **Ovarian Cancer Treatments (Previous Surgeries)**

All the data collected was summarized as the number of previous surgeries (categorically and numerically).

### **Ovarian Cancer Treatments (Previous Systemic Treatments)**

All data collected other than free text was reported: total number of previous lines, total number of each type of treatment received per patient.

## **Progression-Free Survival (PFS)**

PFS: Measured in months from the date of the first dose to the date of the first progression (PD) (whether radiological, clinical or biological) or to the date of death from any cause, whichever occurs first.

### **Objective Response Rate (ORR)**

ORR: Confirmed best overall tumor response of CR or PR according to RECIST v1.1.

### **Adverse Events (AEs)**

The AEs were presented in the summary using counts and frequency percentages. They were stratified by grade and event. The number of events and the number of patients and percentage who had that event was indicated

## **Clinical Laboratory Evaluations**

Laboratory raw variables collected in the baseline visit were summarized.

9.8 Statistical methods

## 9.8.1 Main summary measures

All variables will be summarized separately. Depending on the type of the variable, the following statistics were reported:

- Continuous variables: number of subjects (n), number of missings, mean, standard deviation (STD), median, standard error (SE, if needed), 25th and 75th percentiles, minimum, and maximum.
- Categorical variables: frequencies and percentages (calculated over the number of non-missing values).

In general, minimum and maximum were reported using the same number of decimal places as collected in the raw data. Mean, STD, median, 25th and 75th percentiles will be reported with one additional decimal place.

## 9.8.2 Main statistical methods

Time to event data was listed and summarized at every specified timepoint using the number patients at risk, number of patients censored, number of patients with the event, Kaplan Meier estimate (%), and the 95% confidence interval. In addition, 25th, 50% and 75th percentiles from Kaplan-Meier (KM) curves will be used.

9.8.3 Missing values

No imputation of missing data was performed.

9.8.4 Sensitivity analyses

Not applicable.

9.8.5 Amendments to the statistical analysis plan

No amendments were made to the initial statistical analysis plan.

9.9 Quality control

Each study site was subject to remote clinical monitoring and review by the ethics committees.

The study data was reviewed and cleaned by periodic inspection of the e-CRFs. Remote reviews were performed with enough frequency to ascertain the following:

- Integrity and accuracy of data:
- Informed consent (version, signature and date)

- Eligibility criteria
- e-CRF completion.
- Protocol deviations according GCPs and the applicable regulatory local requirements. Taking appropriate action to prevent recurrence to the detected deviations.
- Compliance with approved protocol and all approved amendments, if any.
- That the investigator receives all documents needed to conduct the study properly and to comply with the applicable regulations.
- That the investigator and local staff are adequately informed about the study through telephone initiation visits.

The study appointed CRO reviewed the e-CRFs for compliance with the protocol, and for inconsistent or missing data. When any missing data or data anomalies were found, queries were sent to the relevant center for resolution. Following the required reviews, the e-CRF data items were exported into the clinical study database for statistical analysis.

# 10. Results

# 10.1 Participants

The study recruited a total of 43 eligible participants.

# 10.2 Descriptive data

Table 1. Subject Disposition. Descriptive Statistics.
All Patients.

| | Total<br>(n=46) |
|-------------------------------------|-----------------|
| Signed Informed Consent | |
| Yes | 46 (100.0%) |
| No | 0 ( 0.0%) |
| Way of signature | |
| Present | 5 ( 10.9%) |
| Absent (definitive) | 41 ( 89.1%) |
| Absent (temporal, by phone) | 0 ( 0.0%) |
| Enrolled patients | |
| Yes | 43 ( 93.5%) |
| No | 3 ( 6.5%) |
| Wavers? | |
| Yes | 0 ( 0.0%) |
| No | 46 (100.0%) |
| Initial Dose of Trabectedin (mg/m2) | |
| N | 43 |
| N Miss | 3 ( 6.5%) |
| Mean | 1.1 |
| Std Dev | 0.1 |
| Median | 1.1 |
| q1 | 1.1 |
| q3 | 1.1 |
| Minimum | 0.8 |
| Maximum | 1.5 |
| Trabectedin split | |
| Missing | 1 ( 2.3%) |
| <1.1 | 7 ( 16.3%) |
| 1.1 | 33 ( 76.7%) |
| >1.1 | 2 ( 4.7%) |

<sup>\*</sup>Trabectedin and PLD initial dose based on patient.

Table 1. Subject Disposition. Descriptive Statistics.
All Patients.

| | Total |
|-----------------------------|-------------|
| | (n=46) |
| Initial Dose of PLD (mg/m2) | |
| N | 43 |
| N Miss | 3 ( 6.5%) |
| Mean | 29.4 |
| Std Dev | 3.3 |
| Median | 30.0 |
| q1 | 30.0 |
| q3 | 30.0 |
| Minimum | 23 |
| Maximum | 46 |
| PLD split | |
| Missing | 1 ( 2.3%) |
| <30 | 8 ( 18.6%) |
| 30 | 33 ( 76.7%) |
| >30 | 1 ( 2.3%) |
| End of treatment | |
| Yes | 44 (100.0%) |
| No | 0 ( 0.0%) |
| Reason of EoT | |
| Patient's decision | 3 ( 6.8%) |
| Doctor's decision | 10 ( 22.7%) |
| Progression | 18 ( 40.9%) |
| Toxicity | 10 ( 22.7%) |
| Other | 3 ( 6.8%) |
| Last Status | - 4 113 |
| Alive with disease | 7 ( 15.9%) |
| Alive without disease | 1 ( 2.3%) |
| Lost to follow-up | 0 ( 0.0%) |
| Dead | 36 ( 81.8%) |
| Progression | 40 ( 05 5%) |
| Yes | 42 ( 95.5%) |
| No | 2 ( 4.5%) |
| Death | 20 / 00 75) |
| Yes | 36 ( 83.7%) |
| No | 7 ( 16.3%) |

<sup>\*</sup>Trabectedin and PLD initial dose based on patient.

Table 1. Subject Disposition. Descriptive Statistics.
All Patients.

| | Total<br>(n=46) |
|--------------------------------|-----------------|
| Reason of Death Ovarian cancer | 35 ( 97.2%) |
| Toxicity | 0 ( 0.0%) |
| Unknown | 1 ( 2.8%) |
| Other | 0 ( 0.0%) |

<sup>\*</sup>Trabectedin and PLD initial dose based on patient.

Table 2. Analysis Sets. Descriptive Statistics.
All Patients.

| | Total |
|--------------------------|-------------|
| | (n=46) |
| Patients with signed ICF | |
| Yes | 46 (100.0%) |
| No | 0 ( 0.0%) |
| Intent-to-Treat | |
| Yes | 43 ( 93.5%) |
| No | 3 ( 6.5%) |
| Safety Analysis Set | |
| Yes | 43 ( 93.5%) |
| No | 3 ( 6.5%) |
| Full Analysis Set | |
| Yes | 43 ( 93.5%) |
| No | 3 ( 6.5%) |
| Per Protocol | |
| Yes | 43 ( 93.5%) |
| No | 3 ( 6.5%) |

Table 3. Patients Characteristics. Descriptive Statistics. Intention to Treat.

| | Total<br>(n=43) |
|----------------------------------------------|-----------------|
| Age (at trabectedin+PLD treatment initiation | |
| according to SmPC) | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 74.7 |
| Std Dev | 3.5 |
| Median | 74.0 |
| q1 | 72.0 |
| q3 | 77.0 |
| Minimum | 70 |
| Maximum | 86 |
| Age | |
| Missing | 0 ( 0.0%) |
| <70 | 0 ( 0.0%) |
| [70-75] | 30 ( 69.8%) |
| >75 | 13 ( 30.2%) |
| Race | |
| White | 41 ( 95.3%) |
| Black or African American | 0 ( 0.0%) |
| Asian | 0 ( 0.0%) |
| American Indian or Alaska Native | 0 ( 0.0%) |
| Native Hawaiian or Other Pacific Islander | 0 ( 0.0%) |
| Unknown | 2 ( 4.7%) |
| Existence of measurable disease | |
| Yes | 35 ( 83.3%) |
| No | 7 ( 16.7%) |
| Existence of bulky disease | |
| Yes | 12 ( 29.3%) |
| No | 29 ( 70.7%) |

Table 3. Patients Characteristics. Descriptive Statistics.
Intention to Treat.

| | Total |
|-----------------------------------------|--------------------------|
| | (n=43) |
| Unight | |
| Weight | 27 |
| N<br>N Mino | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 69.5 |
| Std Dev | 12.2 |
| Median | 69.0 |
| q1 | 59.0 |
| q3 | 79.0 |
| Minimum | 49 |
| Maximum | 94 |
| Weight (Kg) | |
| Missing | 6 ( 14.0%) |
| <58 | 7 ( 16.3%) |
| [58-77] | 18 ( 41.9%) |
| >77 | 12 ( 27.9%) |
| EC OG | |
| 0 | 14 ( 34.1%) |
| 1 | 17 ( 41.5%) |
| 2 | 4 ( 9.8%) |
| 3 | 0 ( 0.0%) |
| 4 | 0 ( 0.0%) |
| Unknown | 6 ( 14.6%) |
| 71-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1- | |
| Platelet count (cells/uL) | 0 ( ( 0 0 0 )) |
| Missing | 6 ( 14.0%) |
| <150000 | 3 ( 7.0%) |
| >-150000 | 34 ( 79.1%) |
| Leukocytes count (10^9/L) | |
| Missing | 6 ( 14.0%) |
| <4500 | 37 ( 86.0%) |
| >-4500 | 0 ( 0.0%) |
| Neutrophils count (cells/uL) | |
| Missing | 6 ( 14.0%) |
| <1500 | 0 ( 0.0%) |
| >-1500 | 37 ( 86.0%) |
| | 5. ( 66.0 <sub>M</sub> / |

Table 3. Patients Characteristics. Descriptive Statistics. Intention to Treat.

| Total<br>(n=43) |
|-------------------------|
| Hemoglobin count (g/dL) |
| Missing 4 ( 9.3%) |
| <11.6 14 ( 32.6%) |
| >-11.6 25 ( 58.1%) |
| CA 125 (U/mL) |
| Missing 6 (14.0%) |
| <-46 5 ( 11.6%) |
| [46-500] 22 ( 51.2%) |
| [500-1000] 7 ( 16.3%) |
| >1000 3 ( 7.0%) |

Table 4. Exposure. Descriptive Statistics.
Intention to Treat.

| | Total<br>(n=43) |
|-------------------------------------|-----------------|
| Initial Dose of Trabectedin (mg/m2) | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 1.1 |
| Std Dev | 0.1 |
| Median | 1.1 |
| q1 | 1.1 |
| q3 | 1.1 |
| Minimum | 0.8 |
| Maximum | 1.5 |
| Trabectedin split | |
| Missing | 1 ( 2.3%) |
| <1.1 | 7 ( 16.3%) |
| 1.1 | 33 ( 76.7%) |
| >1.1 | 2 ( 4.7%) |
| Total dose Trabectedin | |
| N | 35 |
| N Miss | 8 ( 18.6%) |
| Mean | 2.5 |
| Std Dev | 4.4 |
| Median | 1.8 |
| q1 | 1.5 |
| q3 | 1.9 |
| Minimum | 1 |
| Maximum | 28 |
| Initial Dose of PLD (mg/m2) | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 29.4 |
| Std Dev | 3.3 |
| Median | 30.0 |
| q1 | 30.0 |
| q3 | 30.0 |
| Minimum | 23 |
| Maximum | 46 |

Table 4. Exposure. Descriptive Statistics.
Intention to Treat.

| | Total<br>(n=43) |
|--------------------------------|-----------------|
| PLD split | |
| Missing | 1 ( 2.3%) |
| <30 | 8 ( 18.6%) |
| 30 | 33 ( 76.7%) |
| >30 | 1 ( 2.3%) |
| Total dose PLD | |
| N | 35 |
| N Miss | 8 ( 18.6%) |
| Mean | 71.4 |
| Std Dev | 138.2 |
| Median | 49.5 |
| q1 | 42.4 |
| q3 | 53.0 |
| Minimum | 34 |
| Maximum | 865 |
| Duration of treatment (months) | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 4.2 |
| Std Dev | 3.5 |
| Median | 4.0 |
| q1 | 2.0 |
| q3 | 6.0 |
| Minimum | 0 |
| Maximum | 21 |
| Number of cycles | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 5.4 |
| Std Dev | 3.6 |
| Median | 5.0 |
| q1 | 3.0 |
| q3 | 6.0 |
| Minimum | 1 |
| Maximum | 21 |

Table 4. Exposure. Descriptive Statistics.
Intention to Treat.

| | Total (n=43) |
|-------------------------|--------------|
| Number of Cycles | |
| 0 | 0 ( 0.0%) |
| 1 | 2 ( 4.7%) |
| 2 | 8 ( 18.6%) |
| 3 | 6 ( 14.0%) |
| 4 | 3 ( 7.0%) |
| 5 | 3 ( 7.0%) |
| 6 | 11 ( 25.6%) |
| 7 | 1 ( 2.3%) |
| 8 | 3 ( 7.0%) |
| 9 | 1 ( 2.3%) |
| >9 | 5 ( 11.6%) |
| Line of treatment | |
| 2 | 15 ( 34.9%) |
| 3 | 16 ( 37.2%) |
| 4 | 8 ( 18.6%) |
| 5 | 3 ( 7.0%) |
| 6 | 1 ( 2.3%) |
| Number of Interruptions | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 0.0 |
| Std Dev | 0.2 |
| Median | 0.0 |
| q1 | 0.0 |
| q3 | 0.0 |
| Minimum | 0 |
| Maximum | 1 |
| Interruptions | |
| 0 | 42 ( 97.7%) |
| 1 | 1 ( 2.3%) |
| >1 | 0 ( 0.0%) |

Table 4. Exposure. Descriptive Statistics.
Intention to Treat.

| | Total<br>(n=43) |
|-----------------------------|-----------------|
| Fotal days of Interruptions | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 0.0 |
| Std Dev | 0.0 |
| Median | 0.0 |
| q1 | 0.0 |
| q3 | 0.0 |
| Minimum | 0 |
| Maximum | 0 |
| Number of Delayed | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 1.3 |
| Std Dev | 1.5 |
| Median | 1.0 |
| q1 | 0.0 |
| q3 | 2.0 |
| Minimum | 0 |
| Maximum | 7 |
| Delays | |
| 0 | 20 ( 46.5%) |
| 1 | 7 ( 16.3%) |
| 2-4 | 15 ( 34.9%) |
| 5 | 0 ( 0.0%) |
| 6 | 0 ( 0.0%) |
| 7 | 1 ( 2.3%) |
| >7 | 0 ( 0.0%) |
| Total days delated | |
| N | 42 |
| N Miss | 1 ( 2.3%) |
| Mean | 12.3 |
| Std Dev | 15.5 |
| Median | 6.5 |
| q1 | 0.0 |
| q3 | 22.0 |
| Minimum | 0 |
| Maximum | 54 |

Table 4. Exposure. Descriptive Statistics.
Intention to Treat.

| | Total<br>(n=43) |
|--------------------------|-----------------|
| End of treatment | |
| Yes | 43 (100.0%) |
| No | 0 ( 0.0%) |
| Reason of EoT | |
| Patient's decision | 3 ( 7.0%) |
| Doctor's decision | 10 ( 23.3%) |
| Progression | 17 ( 39.5%) |
| Toxicity | 10 ( 23.3%) |
| Other | 3 ( 7.0%) |
| Specify other reason | |
| Infection | 1 ( 33.3%) |
| Knee prothesis infection | 1 ( 33.3%) |
| Unknown | 1 ( 33.3%) |

Listing 1. Duration of Trabectedin + PLD Treatment. Intention to Treat.

\_\_\_\_\_\_ Subjid Site EoT Interruptions Reductions Drugs Exposure 01-001 HUB Yes 0 1 01-002 HUB Yes 0 1 02-001 HRYC Yes 0 1 02-002 HRYC Yes 0 2 3.50 6.13 0.97 3.43 03-001 ICOG Yes 0 2 3.63 03-002 ICOG Yes 3.90 0 2 04-001 HLEO Yes 04-002 HLEO Yes 04-003 HLEO Yes 1 7.00 1 0 0 8.23 0 0 8.70 04-004 HLEO Yes 0 2 4.47 04-005 HLEO Yes 0 0 2.50 04-006 HLEO Yes 0 1 1.20 04-007 HLEO Yes 0 0 1.50 04-008 HLEO Yes 0 2 9.60 05-002 HURS Yes 05-003 HURS Yes 0 0 0.73 0 0 4.70 0 05-004 HURS Yes 0 3.10 0 05-006 HURS Yes 0 4.27 06-001 HCSC Yes 0 0 0.03 06-002 HCSC Yes 0 0 2.13 06-003 HCSC Yes 0 0 1.43 06-004 HCSC Yes 1 0 4.23 06-005 HCSC Yes 06-006 HCSC Yes 0 0 0.77 0 1 5.87 06-007 HCSC Yes 0 0 7.47 06-009 HCSC Yes 0 2 4.37 07-001 HUBA Yes 0 0 1.90 09-001 HUJF Yes 0 0 4.60 09-002 HUJF Yes 0 0 4.00 09-003 HUJF Yes 0 0 1.20 10-001 HVAL Yes 0 1 2.63 0 0 10-002 HVAL Yes 0.03 0 0 10-003 HVAL Yes 7.40 11-001 IVOG Yes 0 0 1.13 11-002 IVOG Yes 0 1 5.67 12-001 HUVR Yes 1 0 1.50 12-002 HUVR Yes 0 1 5.27 12-003 HUVR Yes 12-004 HUVR Yes 0 5.00 1 0 1 0.73 0 20.93 13-001 HVVA Yes 1 14-001 HCVA Yes 0 2 4.23 15-001 HUDP Yes 0

Exposure to Trabectedin+PDL in months

Only patients who have finished treatment (n = 43)

\_\_\_\_\_\_

Listing 1. Duration of Trabectedin + PLD Treatment. Intention to Treat.

| | Subjid |
|---------------------|--------|
| 15-002 HUDP Yes 0 1 | 15-002 |

Exposure to Trabectedin+PDL in months
Only patients who have finished treatment (n = 43)

Table 5. Baseline Laboratory. Descriptive Statistics.
Safetv Analysis Set.

| | Total |
|------------------------------|-------------|
| | (n=43) |
| Platinum sensitivity | |
| Yes | 43 (100.0%) |
| No | 0 ( 0.0%) |
| Platinum-Free Interval (PFI) | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 11.0 |
| Std Dev | 7.2 |
| Median | 9.0 |
| q1 | 7.0 |
| q3 | 11.0 |
| Minimum | 6 |
| Maximum | 42 |
| PFI | |
| Missing | 0 ( 0.0%) |
| 0-10 | 30 ( 69.8%) |
| 11-20 | 11 ( 25.6%) |
| More than 30 | 2 ( 4.7%) |
| Number of previous relapses | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 1.6 |
| Std Dev | 1.0 |
| Median | 1.0 |
| q1 | 1.0 |
| q3 | 2.0 |
| Minimum | 1 |
| Maximum | 5 |
| Previous relapses | |
| Missing | 0 ( 0.0%) |
| 1 | 30 ( 69.8%) |
| 2-3 | 10 ( 23.3%) |
| More than 4 | 3 ( 7.0%) |

Table 5. Baseline Laboratory. Descriptive Statistics. Safety Analysis Set.

| | Total<br>(n=43) |
|---------------------------------|-----------------|
| Progression-Free Survival (PFS) | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 8.3 |
| Std Dev | 8.0 |
| Median | 8.0 |
| q1 | 3.0 |
| q3 | 10.0 |
| Minimum | 0 |
| Maximum | 47 |
| PFS | |
| Missing | 0 ( 0.0%) |
| 0-6 Months | 18 ( 41.9%) |
| 7-12 Months | 18 ( 41.9%) |
| 13-18 Months | 4 ( 9.3%) |
| 19-24 Months | 2 ( 4.7%) |
| 2 Years | 0 ( 0.0%) |
| 3 Years | 1 ( 2.3%) |
| More than 5 Years | 0 ( 0.0%) |
| Weight | |
| N | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 69.5 |
| Std Dev | 12.2 |
| Median | 69.0 |
| q1 | 59.0 |
| q3 | 79.0 |
| Minimum | 49 |
| Maximum | 94 |
| Weight | |
| Missing | 6 ( 14.0%) |
| Less than 40Kg | 0 ( 0.0%) |
| 40-70 Kg | 19 ( 44.2%) |
| 70-100 Kg | 18 (41.9%) |
| More than 100Kg | 0 ( 0.0%) |
| Existence of measurable disease | |
| Yes | 35 ( 81.4%) |
| res<br>No | |
| | 7 ( 16.3%) |
| Missing | 1 ( 2.3%) |
Table 5. Baseline Laboratory. Descriptive Statistics. Safety Analysis Set.

| | Total |
|----------------------------|-------------|
| | (n=43) |
| Existence of bulky disease | |
| Yes | 12 ( 27.9%) |
| No | 29 ( 67.4%) |
| Missing | 2 ( 4.7%) |
| Brain metastasis | |
| Yes | 0 ( 0.0%) |
| No | 43 (100.0%) |
| Platelet count (cells/nL) | |
| N | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 251892 |
| Std Dev | 81702 |
| Median | 241000 |
| q1 | 189000 |
| q3 | 296000 |
| Minimum | 1 2E4 |
| Maximum | 42E4 |
| Platelet count (cells/nL) | |
| Missing | 6 ( 14.0%) |
| Less than 150000 | 3 ( 7.0%) |
| 150000-450000 | 34 ( 79.1%) |
| More than 450000 | 0 ( 0.0%) |
| Leukocytes count (10^9/L) | |
| N | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 6.8 |
| Std Dev | 2.3 |
| Median | 6.5 |
| q1 | 4.9 |
| q3 | 7.7 |
| Minimum | 4 |
| Maximum | 14 |
| Leukocytes count (10^9/L) | |
| Missing | 6 ( 14.0%) |
| Less than 4.5 | 4 ( 9.3%) |
| 4.5-11.0 | 33 ( 76.7%) |
| More than 11.0 | 0 ( 0.0%) |

Table 5. Baseline Laboratory. Descriptive Statistics. Safety Analysis Set.

| | Total<br>(n=43) |
|---------------------------------|-----------------|
| Absolute Neutrophils (cells/nL) | |
| N | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 4148.9 |
| Std Dev | 1812.0 |
| Median | 3820.0 |
| q1 | 3000.0 |
| q3 | 4970.0 |
| Minimum | 1830 |
| Maximum | 8880 |
| Absolute Neutrophils (cells/nL) | |
| Missing | 6 ( 14.0%) |
| Less than 1500 | 0 ( 0.0%) |
| 1500-8000 | 0 ( 0.0%) |
| More than 8000 | 0 ( 0.0%) |
| 1500-80 | 35 ( 81.4%) |
| More th | 2 ( 4.7%) |
| Hemoglobin (g/dL) | |
| N | 39 |
| N Miss | 4 ( 9.3%) |
| Mean | 12.0 |
| Std Dev | 1.5 |
| Median | 12.1 |
| q1 | 11.0 |
| q3 | 13.4 |
| Minimum | 8 |
| Maximum | 15 |
| Hemoglobin (g/dL) | |
| Missing | 4 ( 9.3%) |
| Less than 11.6 | 14 ( 32.6%) |
| 11.6-15.0 | 25 ( 58.1%) |
| More than 15.0 | 0 ( 0.0%) |

Table 5. Baseline Laboratory. Descriptive Statistics.
Safety Analysis Set.

| | Tota | al |
|-----------------|-------|----------|
| | (n=4 | |
| | \II - | .07 |
| (A10E (II/mI) | | |
| CA125 (U/mL) | | |
| N | 37 | |
| N Miss | 6 ( | 14.0%) |
| Mean | 452.1 | |
| Std Dev | 780.4 | <u>l</u> |
| Median | 174.9 | ) |
| q1 | 67.0 | ) |
| q3 | 540.0 | ) |
| Minimum | 0 | |
| Maximum | 4389 | |
| CA125 (U/mL) | | |
| Missing | 6 ( | (14.0%) |
| Less than 46.0 | 5 ( | 11.6%) |
| 46.0-200.0 | 16 ( | (37.2%) |
| More than 200.0 | | 37.2%) |

Table 6. Concomitant Medication. Descriptive Statistics.
Intention to Treat.

Stage Trabectidin+PLD Reason Total \_\_\_\_\_ Before Antiacid SUBJECTS 1 ( 2.3%) EPISODES 1 Prophylaxis Anticoagulant SUBJECTS 1 ( 2.3%) EPISODES 1 Medical history comorbidities Antidepressant SUBJECTS 1 ( 2.3%) EPISODES 1 Medical history comorbidities Antiemetic SUBJECTS 2 ( 4.7%) Prophylaxis EPISODES 2 Antihypertensive Medical history comorbidities SUBJECTS 2 ( 4.7%) EPISODES Colony-stimulating factor SUBJECTS 1 ( 2.3%) EPISODES 1 Adverse event Diuretic SUBJECTS 1 ( 2.3%) EPISODES 1 Other Magnesium (supplement) SUBJECTS 1 ( 2.3%) EPISODES 1 Prophylaxis Proton-pump inhibitor SUBJECTS 1 ( 2.3%) EPISODES 1 Prophylaxis Transfusion SUBJECTS 1 ( 2.3%) Adverse event EPISODES Vitamin B12 (supplement) SUBJECTS 1 ( 2.3%) EPISODES 1 Prophylaxis Other SUBJECTS 1 ( 2.3%) EPISODES 1 Prophylaxis During Antibiotic

Table 6. Concomitant Medication. Descriptive Statistics.
Intention to Treat.

-----

| Stage Trabectidin+PLD Type | | | |
|---------------------------------|----------------------|-------|-------|
| Reason | | Total | |
| Adverse event | SUBJECTS | | 4.7%) |
| 1-4:1:1-1 | EPISODES | 2 | |
| Antidiarrheal medication | CUD IECTO | | 0 247 |
| Adverse event | SUBJECTS<br>EPISODES | 1 | 2.3%) |
| Antiemetic | | | |
| Adverse event | SUBJECTS | 2 ( | 4.7%) |
| | EPISODES | 2 | |
| Antifungal | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Apetite stimulant | | | |
| Other | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Colony-stimulating factor | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Corticosteroid | | | |
| Adverse event | SUBJECTS | 2 ( | 4.7%) |
| | EPISODES | 2 | |
| Potassium chloride (supplement) | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Transfusion | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Other | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Before and During | | | |
| Analgesic | | | |
| Adverse event | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 1 | |
| Other | SUBJECTS | 1 ( | 2.3%) |
| | EPISODES | 2 | |
| Prophylaxis | SUBJECTS | 3 ( | 7.0%) |
| | EPISODES | 3 | |
| Antiacid | | | |
| Prophylaxis | SUBJECTS | 4 ( | 9.3%) |
| | EPISODES | 4 | |

Table 6. Concomitant Medication. Descriptive Statistics.
Intention to Treat.

Stage Trabectidin+PLD

| Stage Trabectidin+PLD | | |
|-----------------------------------|-----------|------------|
| Туре | | |
| Reason | | Total |
| Antibiotic | | |
| Prophylaxis | | 1 ( 2.3%) |
| | EPISODES | 1 |
| Antidepressant | | |
| Medical history comorbidities | SUBJECTS | 4 ( 9.3%) |
| | EPISODES | 4 |
| Prophylaxis | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 2 |
| Antidiabetic medication | | |
| Medical history comorbidities | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 2 |
| Antiemetic | | |
| Adverse event | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Antihistamine | | |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Antihypertensive | | |
| Medical history comorbidities | SUBJECTS | 5 ( 11.6%) |
| • | EPISODES | 5 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Antiplatelet drug (antiaggregant) | | |
| Medical history comorbidities | SUBJECTS | 2 ( 4.7%) |
| • | EPISODES | 2 |
| Benzodiazepines | | |
| Medical history comorbidities | SUBJECTS | 2 ( 4.7%) |
| • | EPISODES | 2 |
| Prophylaxis | SUBJECTS | 3 ( 7.0%) |
| | EPISODES | 3 |
| Colony-stimulating factor | | _ |
| Adverse event | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Corticosteroid | | - |
| Other | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| | 1. 100DH0 | - |

Table 6. Concomitant Medication. Descriptive Statistics.
Intention to Treat.

| Stage Trabectidin+PLD<br>Type | | |
|-------------------------------|----------|------------|
| Reason | | Total |
| Diuretic | | |
| Medical history comorbidities | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Laxative | | |
| Medical history comorbidities | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Magnesium (supplement) | | |
| Medical history comorbidities | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Iron sulfate (supplement) | | |
| Medical history comorbidities | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Proton-pump inhibitor | | |
| Other | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Prophylaxis | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 2 |
| Statins | | |
| Medical history comorbidities | SUBJECTS | 5 ( 11.6%) |
| | EPISODES | 5 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Other | | |
| Adverse event | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Medical history comorbidities | SUBJECTS | 4 ( 9.3%) |
| | EPISODES | 5 |
| Other | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 3 |
| Prophylaxis | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |

------

Listing 2. Concomitant Medication. Intention to Treat.

| Subjid | Site St | age** | Type Med/Therapy* | Reason* |
|---|---|---|---|---|
| 01-001 | HUB | BT | Antidepressant | MHC: Paroxetina |
| | | BDT | Antidiabetic Medication | MHC: Sitagliptina |
| | | DT | Antidiarrheal Medication | AE: Movicol |
| | | BT | Antiemetic | Prophylaxis |
| | | BDT | Statins | MHC: Atorvastatina |
| 01-002 | HUB | DT | Antifungal | AE: Mycostatin |
| | | BT | Antihypertensive | MHC: Enalapril |
| | | BT | Antihypertensive | MHC: Sutril |
| | | BT | Magnesium (Supp) | Prophylaxis |
| | | BT | 0: Orfidal | Prophylaxis |
| | | BT | Proton-Pump Inhibitor | Prophylaxis |
| 02-002 | HRYC | BT | Antiacid | Prophylaxis |
| | | BDT | Antihypertensive | MHC: Hypertension |
| | | DT | Colony-Stimulating Factor | AE: Neutropenia |
| | | BT | Diuretic | O: Hepatotoxicity |
| 03-001 | ICOG | DT | Antibiotic | AE: Urinary Tract Infection |
| | | BDT | Colony-Stimulating Factor | AE: Neutrophil Count Decrease |
| 03-002 | ICOG | DT | Antibiotic | AE: Urinary Tract Infection |
| 04-001 | HLEO | BDT | Analgesic | Prophylaxis |
| | | BDT | Antidepressant | MHC: Depression |
| | | BDT | O: Morphine | O: Pain Disease |
| | | BDT | Statins | MHC: Dislipemia |
| 04-002 | HLEO | BDT | Analgesic | Prophylaxis |
| | | BDT | Antiacid | Prophylaxis |
| | | BDT | Antihypertensive | MHC: Arterial Hypertension |
| | | BDT | Iron Sulfate (Supp) | Prophylaxis |
| | | BDT | Statins | MHC: Dislipemia |
| 04-003 | HLEO | BDT | Antiacid | Prophylaxis |
| | | BDT | Antiemetic | Prophylaxis |
| 04-004 | HLEO | DT | O: Neupogen | AE: Neutropenia |
| 04-005 | HLEO | BDT | Antidiabetic Medication | MHC: Diabetes Mellitus |
| | | BDT | Benzodiazepines | Prophylaxis |
| 04-006 | HLEO | BDT | Antidepressant | Prophylaxis |
| | | BDT | Antihistamine | Prophylaxis |
| | | BDT | Antihypertensive | MHC: Arterial Hipertension |
| | | BDT | Statins | MHC: Dislipemia |
| 04-007 | HLEO | BDT | Antihypertensive | MHC: Arterial Hipertension |
| | | BDT | Benzodiazepines | Prophylaxis |
| | | BDT | Laxative | MHC: Constipation |
| | | BT | Vitamin B12 (Supp) | Prophylaxis |
| 04-008 | HLEO | BDT | Analgesic | Prophylaxis |

<sup>\*\*</sup>BT - Before Treatment, DT - During Treatment, BDT - Before and During treatment

<sup>\*</sup>O - Other, MHC - Medical history comorbidities

<sup>\*</sup>supp = Supplement, AA = Antiaggregant, AE = Adverse Event

Listing 2. Concomitant Medication. Intention to Treat.

| Subjid | Site St | age** | Type Med/Therapy* | Reason* |
|---|---|---|---|---|
| | | BDT | Antiacid | Prophylaxis |
| | | BDT | Benzodiazepines | Prophylaxis |
| | | BDT | Statins | MHC: Dislipemia |
| 05-002 | HURS | DT | Corticosteroid | AE: Nausea And Vomiting |
| 05-003 | HURS | BT | Antihypertensive | MHC: Hypertension |
| | | BDT | O: Potassium | AE: Hypokalemia |
| | | DT | Potassium Chloride (Supp) | AE: Hypokalemia |
| 09-003 | HUJF | DT | Antiemetic | AE: Nausea And Vomiting |
| | | BDT | Diuretic | MHC: Ascites |
| 10-001 | HVAL | BDT | Antiplatelet Drug (Aa) | MHC: Unknown |
| | | BDT | Benzodiazepines | MHC: Anxiety |
| | | BDT | 0: Lipid-Lowering | MHC: Hyperclesterolemia |
| 11-001 | IVOG | BDT | Antihypertensive | MHC: Amlodipino 10mg |
| | | BDT | Antihypertensive | MHC: Bisoprolol 5mg |
| | | BDT | Antihypertensive | MHC: Hidroclorotiazida 12.5mg |
| | | BDT | Antihypertensive | MHC: Valsartán 160mg |
| 11-002 | IVOG | BT | Anticoagulant | MHC: Hibor 10000 Ui |
| 12-002 | HUVR | BDT | O: Levotiroxine | MHC: Hypothyrodism |
| | | BDT | Proton-Pump Inhibitor | Prophylaxis |
| 12-003 | HUVR | BDT | Antidepressant | MHC: Depression |
| | | BDT | Antiemetic | AE: Nausea |
| | | BT | Antiemetic | Prophylaxis |
| | | BDT | Benzodiazepines | MHC: Depression |
| | | BT | Colony-Stimulating Factor | AE: Neutropenia |
| | | BDT | Corticosteroid | O: Intestinal Suboclusion Bt |
| | | BDT | Laxative | Prophylaxis |
| | | BDT | O: Fentanyl (Patch) | O: Intestinal Suboclusion Bt |
| | | BDT | O: Morphine | O: Intestinal Suboclusion Bt |
| | | BDT | Proton-Pump Inhibitor | O: Intestinal Suboclusion Bt |
| | | BT | Transfusion | AE: Anemia |
| 12-004 | HUVR | BDT | Analgesic | O: Cancer-Related Pain |
| | | BDT | Analgesic | O: Cancer-Related Pain |
| | | BDT | Antibiotic | Prophylaxis |
| | | BDT | Antidepressant | MHC: Depression |
| | | DT | Antiemetic | AE: Nausea And Vomiting |
| | | BDT | Antiplatelet Drug (Aa) | MHC: Chronic Leg Ischemya |
| | | DT | Apetite Stimulant | O: Cancer-Related Hyporexia |
| | | DT | Corticosteroid | AE: Asthenia |
| | | BDT | Iron Sulfate (Supp) | MHC: Renal Failure |
| | | BDT | Magnesium (Supp) | MHC: Renal Failure |
| | | BDT | O: Ciclosporine | MHC: Renal Trasplant |
| | | | • | • |

<sup>\*\*</sup>BT - Before Treatment, DT - During Treatment, BDT - Before and During treatment

<sup>\*</sup>O - Other, MHC - Medical history comorbidities

<sup>\*</sup>supp = Supplement, AA = Antiaggregant, AE = Adverse Event

Listing 2. Concomitant Medication. Intention to Treat.

| ıbjid | Site S | tage** | Type Med/Therapy* | Reason* |
|---|---|---|---|---|
| | | BDT | O: Levotiroxine | MHC: Hypothyroidism |
| | | BDT | Proton-Pump Inhibitor | Prophylaxis |
| | | DT | Transfusion | AE: Anemia G2 |
| 13-001 | HVVA | BDT | Antidepressant | Prophylaxis |
| | | BDT | O: Anxiolytic | Prophylaxis |
| 14-001 | HCVA | BDT | Antidepressant | MHC: Depression |
| | | BDT | Antihypertensive | Prophylaxis |
| | | BDT | Diuretic | Prophylaxis |
| | | BDT | Statins | Prophylaxis |
| 15-001 | HUDP | BDT | Analgesic | AE: Abdominal Pain |
| 15-002 | HUDP | BDT | Antiacid | Prophylaxis |
| | | BDT | Corticosteroid | Prophylaxis |
| | | BDT | 0: Thyroideal Hormones | MHC: Total Thyroidectomy In 1982 Fo |

<sup>\*\*</sup>BT - Before Treatment, DT - During Treatment, BDT - Before and During treatment

Table 7. Medical History. Descriptive Statistics.
Intention to Treat.

| | Total<br>(n=43) |
|---------------------------|-----------------|
| Relevant Comorbidities | |
| Yes | 33 ( 76.7%) |
| No | 10 ( 23.3%) |
| Other Previous Cancers | |
| Yes | 6 ( 14.0%) |
| No | 37 ( 86.0%) |
| Family history of Cancers | |
| Yes | 30 ( 69.8%) |
| No | 13 ( 30.2%) |

<sup>\*</sup>O - Other, MHC - Medical history comorbidities

<sup>\*</sup>supp = Supplement, AA = Antiaggregant, AE = Adverse Event

Table 7.1. Medical History. Descriptive Statistics.
Intention to Treat.

| | Total |
|-------------------------------|-------------|
| | (n=43) |
| amily history of Cancers | |
| Yes | 30 ( 69.8%) |
| No | 13 ( 30.2%) |
| Familiars with cancer | |
| Aunt | 6 ( 10.0%) |
| Brother | 11 ( 18.3%) |
| Cousin | 7 ( 11.7%) |
| Daughter | 1 ( 1.7%) |
| Father | 9 ( 15.0%) |
| Grandchild | 1 ( 1.7%) |
| Grandfather | 1 ( 1.7%) |
| Grandmother | 2 ( 3.3%) |
| Mother | 7 ( 11.7%) |
| Niece | 1 ( 1.7%) |
| None | 1 ( 1.7%) |
| Sister | 9 (15.0%) |
| Uncle | 4 ( 6.7%) |
| Types of cancer<br>Bile Ducts | 1 ( 1.7%) |
| Bladder | 1 ( 1.7%) |
| Breast | 14 ( 23.3%) |
| Colon | 7 ( 11.7%) |
| Esophagus | 1 ( 1.7%) |
| Gallbladder | 1 ( 1.7%) |
| Gastric | 6 ( 10.0%) |
| Hepatocarcinoma | 1 ( 1.7%) |
| Kaposi Sarcoma | 1 ( 1.7%) |
| Liver | 3 ( 5.0%) |
| Lung | 3 ( 5.0%) |
| None | 1 ( 1.7%) |
| Ovarian | 2 ( 3.3%) |
| Pancreas | 6 ( 10.0%) |
| Parotide | 1 ( 1.7%) |
| Prostate | 4 ( 6.7%) |
| Renal | 1 ( 1.7%) |
| Testicles | 1 ( 1.7%) |
| Unknown | 3 ( 5.0%) |
| Uterine | 2 ( 3.3%) |

Listing 3. Medical History. Family History of Cancers. Intention to Treat. Intention to Treat.

| | Site C | ancer in Family | Member | Туре |
|--------|--------|-----------------|---------------|-----------------|
| | HUB | | Brother | Lung |
| | | | Cousin | Gastric |
| 01-002 | HUB | Yes | Mother | Breast |
| | | | Brother | Gastric |
| | HRYC | | | |
| 02-002 | HRYC | Yes | Mother | Pancreas |
| | | | Brother | O: Bile Ducts |
| | | | Uncle | Gastric |
| | | | Cousin | Breast |
| | | | Aunt | Pancreas |
| 03-001 | ICOG | No | | |
| 03-002 | ICOG | Yes | Brother | Prostate |
| | | | Brother | Unknown |
| 04-001 | HLEO | Yes | 0: Grandchild | Testicles |
| | | | Brother | Colon |
| 04-002 | HLEO | Yes | Sister | Breast |
| | | | Sister | Colon |
| | | | Brother | O: Renal |
| 04-003 | HLEO | No | | |
| 04-004 | HLEO | Yes | Grandmother | Unknown |
| 04-005 | HLEO | No | | |
| 04-006 | HLEO | Yes | Brother | Liver |
| | | | Brother | Liver |
| 04-007 | HLEO | Yes | Sister | Breast |
| | | | Father | Pancreas |
| | | | O: Niece | Breast |
| 04-008 | HLEO | Yes | 0: Daughter | Ovarian |
| 05-002 | HURS | Yes | Mother | Breast |
| | | | Aunt | Breast |
| | | | Cousin | Breast |
| 05-003 | HURS | No | | |
| 05-004 | HURS | No | | |
| 05-006 | HURS | No | | |
| 06-001 | HC SC | Yes | Brother | Colon |
| 06-002 | HC SC | Yes | Father | Prostate |
| | | | Uncle | Prostate |
| | | | Uncle | Prostate |
| | | | Uncle | O: Hepatocarcin |
| 06-003 | HC SC | No | | • |
| 06-004 | HCSC | | | |

\*0 - Other

Listing 3. Medical History. Family History of Cancers. Intention to Treat. Intention to Treat.

| Subjid | Site | Cancer | in Family | Member | Туре |
|--------|------|--------|-----------|-------------|-----------------|
| 06-005 | HC S | C Yes | | Father | Colon |
| | | | | Aunt | 0: Pancreas |
| | | | | Grandmother | O: Pancreas |
| | | | | Aunt | Breast |
| | | | | Aunt | Colon |
| | | | | Cousin | Breast |
| 06-006 | HCS | C Yes | | Father | Colon |
| | | | | Aunt | Breast |
| | | | | Mother | O: Kaposi Sarco |
| 06-007 | HCS | C Yes | | Grandfather | O: Parotide |
| | | | | Cousin | Uterine |
| | | | | Cousin | 0: Bladder |
| 06-009 | HCS | C Yes | | Father | 0: Esophagus |
| 07-001 | HUB | A Yes | | Sister | Colon |
| 09-001 | HUJ | F Yes | | Mother | Liver |
| | | | | Father | Unknown |
| | | | | Sister | Uterine |
| 09-002 | HUJ | F Yes | | Brother | Lung |
| 09-003 | HUJ | F No | | | |
| 10-001 | HVA | L Yes | | Sister | Breast |
| 10-002 | HVA | L Yes | | Cousin | Breast |
| 10-003 | HVA | L Yes | | Sister | Ovarian |
| 11-001 | IVO | G No | | | |
| 11-002 | IVO | G No | | | |
| 12-001 | HUV | R Yes | | Mother | 0: Gallbladder |
| | | | | Father | Lung |
| 12-002 | HUV | R Yes | | Father | Gastric |
| 12-003 | HUV | R Yes | | Father | Gastric |
| 12-004 | HUV | R No | | | |
| 13-001 | HVV | A Yes | | Sister | Breast |
| 14-001 | HCV | A Yes | | Sister | Gastric |
| 15-001 | HUD | P Yes | | Mother | Pancreas |
| 15-002 | HUD | P Yes | | O: None | O: None |

\*0 - Other

Table 7.2. Medical History. Other Previous Cancers. Descriptive Statistics. Intention to Treat.

| | Total<br>(n=43) |
|-----------------------------|-----------------|
| Previous Cancers | |
| Yes | 6 ( 14.0%) |
| No | 37 ( 86.0%) |
| Cancer Type | |
| Breast | 3 ( 50.0%) |
| Carcinoid Tumor in Appendix | 1 ( 16.7%) |
| Peritoneal Carcinomatosis | 1 ( 16.7%) |
| Thyroideal Cancer | 1 ( 16.7%) |

Listing 4. Medical History. Family History of Cancers.

| Subjid | Site Pr | evious Cancer | Cancer type |
|--------|----------------|---------------|------------------------------|
| - | | | |
| | HUB | | |
| 01-002 | HUB<br>HRYC | Yes | Breast |
| 02-001 | HRYC | No | |
| | HRYC | | |
| 03-001 | ICOG | No | |
| 03-002 | ICOG<br>HLEO | No | |
| | | | 0: Peritoneal Carcinomatosis |
| | HLEO | | |
| 04-003 | HLEO<br>HLEO | No | |
| 04-004 | HLEO | Yes | Carcinoid Tumor in Appendix |
| | HLEO | | |
| 04-006 | HLEO | No | |
| 04-007 | HLEO<br>HLEO | No | |
| | | | Breast |
| | HURS | | |
| 05-003 | HURS | No | |
| 05-004 | HURS | No | |
| | HURS | | |
| | HC SC | No | |
| 06-002 | HC SC<br>HC SC | No | |
| | HCSC | | |
| 06-005 | HC SC<br>HC SC | No | |
| 06-006 | HC SC | No | |
| | HCSC | | |
| 06-009 | HC SC | No | |
| 07-001 | HUBA<br>HUJF | No | |
| | HUJF | | |
| 09-003 | HUJF | Yes | Breast |
| 10-001 | HVAL | No | |
| | HVAL | | |
| | HVAL | | |
| 11-001 | IVOG<br>IVOG | No | |
| | HUVR | | |
| 12-002 | HUVR | No | |
| 12-003 | HUVR | No | |
| | HUVR | | |
| 13-001 | HVVA | NO | |

\*0 - Other

Listing 4. Medical History. Family History of Cancers.

| Subjid | Site Pr | evious Cancer | Cancer type |
|---|---|---|---|
| 14-001<br>15-001<br>15-002 | HCVA<br>HUDP<br>HUDP | No<br>No<br>Yes | O: Thyroideal Cancer |
| *0 - Other | <br>r | | |

Table 7.3. Medical History. Relevant Comorbidities. Descriptive Statistics.

| | Total |
|--------------------------|-------------|
| | (n=43) |
| | (11-45) |
| Relevant Comorbidities | |
| No | 10 ( 23.3%) |
| Yes | 33 ( 76.7%) |
| Time point | |
| Baseline | 7 ( 8.3%) |
| Medical History | 77 ( 91.7%) |
| | ( 52,/ |
| Relevant comorbidities | |
| Anxiety | 1 ( 1.2%) |
| • | 18 ( 21.4%) |
| Arterial hypertension | |
| Arthrosis | 1 ( 1.2%) |
| COPD | 1 ( 1.2%) |
| Cerebrovascular disease | 1 ( 1.2%) |
| Depression | 8 ( 9.5%) |
| Diabetes mellitus | 4 ( 4.8%) |
| Dyslipemia | 13 ( 15.5%) |
| Hypothiroidism | 3 ( 3.6%) |
| Obesity | 1 ( 1.2%) |
| Other relevant (Specify) | 33 ( 39.3%) |

Table 7.3. Medical History. Relevant Comorbidities. Descriptive Statistics.

Total (n=43)Specify Allergy To Clavulanic Acid 1 ( 3.0%) 1 ( 3.0%) Anal Fissure 1 ( 3.0%) Appendectomy 1 ( 3.0%) Ascites Atrial Fibrillation 1 ( 3.0%) Carpal Tunnel Surgery 1 ( 3.0%) Chronic Leg Ischemya 1 ( 3.0%) Chronic Renal Disease 2 ( 6.1%) 1 ( 3.0%) Colecistectomy 1 ( 3.0%) Constipation 1 ( 3.0%) Cured Hepatitis B 1 ( 3.0%) Curettage Deep Vein Thrombosis 1 ( 3.0%) Finger Amputation 1 ( 3.0%) Goitre 1 ( 3.0%) Hernia 4 ( 12.1%) Internal Hemorrhoids 1 ( 3.0%) 1 ( 3.0%) Lichen Planus 1 ( 3.0%) Lipoma Surgery In Left Arm Osteoporosis 3 ( 9.1%) Parietotemporal Hematoma Surgery 1 ( 3.0%) Peripheral Neuropathy 1 ( 3.0%) Polymyalgia Rheumatica 1 ( 3.0%) 1 ( 3.0%) Tendinopathy Tibial Plateau Fracture 1 ( 3.0%) 1 ( 3.0%) Varicose Veins Vertiginous Syndrome 1 ( 3.0%)

\_\_\_\_\_\_

Listing 5. Medical History. Relevant Comorbidities. Intention to Treat.

| MH Dyslipemia MH D: Peripheral Neuropathy MH Depression MH Depression MH O: Carpal Tunnel Surgery O4-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-003 HLEO Yes MH Dyslipemia O4-004 HLEO Yes MH Dyslipemia O5 Tibial Plateau Fracture MH Depression MH Depression O6 Finger Amputation O4-005 HLEO Yes MH Diabetes Mellitus O4-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | Time<br>Subjid | Site C | omorbidities | point | Туре |
|---|---|---|---|---|---|
| BL Diabetes Mellitus MH Arterial Hypertension MH O: Bocio MH O: Osteoporosis O2-001 HRYC No O2-002 HRYC Yes MH Arterial Hypertension MH Copd MH O: Osteoporosis MH O: Internal Hemorrhoids O3-001 ICOG Yes MH Arterial Hypertension MH Depression MH Depression MH Hypothiroidism O4-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH O: Peripheral Neuropathy MH Depression MH Dyslipemia O4-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-003 HLEO Yes MH O: Hernia MH Arterial Hypertension O4-004 HLEO Yes MH Diabetes Mellitus O4-005 HLEO Yes MH Diabetes Mellitus O4-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-007 HLEO Yes MH Arterial Hypertension MH Diabetes Mellitus O4-007 HLEO Yes MH Arterial Hypertension MH Diabetes Mellitus O5 Pinger Amputation MH Dyslipemia O6 Vertiginous Syndrome MH O: Vertiginous Syndrome MH O: Hernia MH O: Hernia MH O: Hernia MH O: Hernia MH O: Hernia MH O: Hernia | 01-001 | HUB | Yes | МН | Dyslipemia |
| O1-002 | | | | MH | Depression |
| MH | | | | BL | Diabetes Mellitus |
| MH | 01-002 | HUB | Yes | MH | Arterial Hypertension |
| O2-002 | | | | MH | O: Bocio |
| O2-002 | | | | MH | O: Osteoporosis |
| MH | 02-001 | HRYC | No | | |
| MH | 02-002 | HRYC | Yes | MH | Arterial Hypertension |
| MH O: Internal Hemorrhoids 03-001 ICOG Yes MH Arterial Hypertension 03-002 ICOG Yes MH Arterial Hypertension MH Depression MH Hypothiroidism 04-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH Depression MH Depression MH Depression MH Depression MH Depression MH Dyslipemia 0: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-004 HLEO Yes MH O: Hernia MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia MH O: Tibial Plateau Fracture MH Depression MH O: Finger Amputation 04-006 HLEO Yes MH Arterial Hypertension 04-006 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH Arterial Hypertension MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia MH O: Hernia | | | | MH | • |
| 03-001 ICOG Yes MH Arterial Hypertension 03-002 ICOG Yes MH Arterial Hypertension 04-001 HLEO Yes MH Depression MH Dyslipemia MH Depression MH Depression MH Depression MH Depression MH Depression MH Dyslipemia MH Dyslipemia 04-003 HLEO Yes MH Dyslipemia 04-004 HLEO Yes MH Dyslipemia 04-004 HLEO Yes MH Diabetes Mellitus 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH O: Vertiginous Syndrome 04-007 HLEO Yes MH O: Vertiginous Syndrome 04-007 HLEO Yes MH O: Hernia 04-007 | | | | MH | O: Osteoporosis |
| O3-002 ICOG Yes MH Arterial Hypertension MH Depression MH Hypothiroidism O4-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH Depression MH Depression MH Depression MH Depression MH O: Carpal Tunnel Surgery O4-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-003 HLEO Yes MH O: Hernia MH Arterial Hypertension O4-004 HLEO Yes MH Dyslipemia O4-005 HLEO Yes MH Depression O4-005 HLEO Yes MH Diabetes Mellitus O4-006 HLEO Yes MH Diabetes Mellitus O4-007 HLEO Yes MH O: Vertiginous Syndrome MH Dyslipemia O4-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia MH O: Hernia | | | | MH | 0: Internal Hemorrhoids |
| MH Depression MH Hypothiroidism 04-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH Depression MH Depression MH Depression MH Depression MH Depression MH Depression MH Dyslipemia 04-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-003 HLEO Yes MH O: Hernia MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia MH Depression MH Depression MH Depression MH Depression MH Depression MH Depression MH Diabetes Mellitus 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH D: Constipation MH Arterial Hypertension MH Arterial Hypertension MH Arterial Hypertension MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia | 03-001 | ICOG | Yes | MH | |
| MH Hypothiroidism 04-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH O: Peripheral Neuropathy MH Depression MH O: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-003 HLEO Yes MH O: Hernia MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Depression MH O: Tibial Plateau Fracture MH Depression MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | 03-002 | ICOG | Yes | MH | Arterial Hypertension |
| 04-001 HLEO Yes MH O: Allergy To Clavulanic Aci MH Dyslipemia MH O: Peripheral Neuropathy MH Depression MH O: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-003 HLEO Yes MH O: Hernia MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Depression 04-006 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Constipation MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia MH O: Hernia | | | | MH | • |
| MH Dyslipemia MH D: Peripheral Neuropathy MH Depression MH Depression MH O: Carpal Tunnel Surgery O4-002 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-003 HLEO Yes MH Dyslipemia O4-004 HLEO Yes MH Dyslipemia O5 Tibial Plateau Fracture MH Depression MH Depression O6-005 HLEO Yes MH Diabetes Mellitus O4-006 HLEO Yes MH Arterial Hypertension O4-007 HLEO Yes MH Arterial Hypertension MH Dyslipemia O4-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | Hypothiroidism |
| MH O: Peripheral Neuropathy MH Depression MH O: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension 04-003 HLEO Yes MH O: Hernia 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Depression 04-006 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH O: Vertiginous Syndrome 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | 04-001 | HLEO | Yes | MH | O: Allergy To Clavulanic Acid |
| MH Depression MH O: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension 04-003 HLEO Yes MH O: Hernia 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH Dyslipemia 04-007 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH Dyslipemia 04-007 HLEO Yes MH Dyslipemia 05 Vertiginous Syndrome 06 Constipation MH O: Constipation MH Arterial Hypertension MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | Dyslipemia |
| MH O: Carpal Tunnel Surgery 04-002 HLEO Yes MH Arterial Hypertension 04-003 HLEO Yes MH O: Hernia 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Depression 04-006 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia MH O: Hernia | | | | MH | |
| 04-002 HLEO Yes MH Arterial Hypertension 04-003 HLEO Yes MH O: Hernia 04-004 HLEO Yes MH Dyslipemia 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Depression 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH O: Vertiginous Syndrome 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | - |
| MH Dyslipemia 04-003 HLEO Yes MH O: Hernia MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia MH Depression MH Depression MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH O: Hernia MH O: Hernia MH O: Hernia | | | | | |
| 04-003 HLEO Yes MH O: Hernia 04-004 HLEO Yes MH Dyslipemia 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension 04-007 HLEO Yes MH Diabetes Mellitus 04-007 HLEO Yes MH O: Vertiginous Syndrome 04-007 MH O: Constipation MH O: Hernia MH O: Hernia MH O: Hernia | 04-002 | HLEO | Yes | MH | |
| MH Arterial Hypertension 04-004 HLEO Yes MH Dyslipemia MH Depression MH Depression MH Diabetes Mellitus 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH D: Constipation MH D: Hernia MH O: Hernia | | | | MH | |
| 04-004 HLEO Yes MH Dyslipemia MH D: Tibial Plateau Fracture MH Depression MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia | 04-003 | HLEO | Yes | MH | |
| MH O: Tibial Plateau Fracture MH Depression MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | | |
| MH Depression MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | 04-004 | HLEO | Yes | | <i>y</i> 1 |
| MH O: Finger Amputation 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | |
| 04-005 HLEO Yes MH Diabetes Mellitus 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | - |
| 04-006 HLEO Yes MH Arterial Hypertension MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | MH | · . |
| MH Dyslipemia 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | 04-005 | | | MH | |
| 04-007 HLEO Yes MH O: Vertiginous Syndrome MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | 04-006 | HLEO | Yes | MH | 0.1 |
| MH O: Constipation MH Arterial Hypertension MH O: Hernia MH O: Hernia | | | | | |
| MH Arterial Hypertension<br>MH O: Hernia<br>MH O: Hernia | 04-007 | HLEO | Yes | | |
| MH O: Hernia<br>MH O: Hernia | | | | | • |
| MH 0: Hernia | | | | | |
| MH Π: Linoma Surgery In Left Δτ | | | | | |
| | | | | MH | O: Lipoma Surgery In Left Arm |
| MH O: Curettage | | | | | _ |
| 04-008 HLEO Yes MH Diabetes Mellitus | 04-008 | HLEO | Yes | | |
| MH Dyslipemia | | | | MH | Dyslipemia |

<sup>\*0 -</sup> Other

<sup>\*</sup>MH - Medical History, BL - Baseline

Listing 5. Medical History. Relevant Comorbidities. Intention to Treat.

\_\_\_\_\_ Time Subjid Site Comorbidities point Type \_\_\_\_\_ 05-002 HURS Yes MH Diabetes Mellitus Dyslipemia MH 05-003 HURS Yes Arterial Hypertension MH MH 0: Hernia MH 0: Anal Fissure MH 0: Colecistectomy
MH 0: Appendectomy
MH 0: Tendonitis 05-004 HURS No 05-006 HURS No 06-001 HCSC No 06-002 HCSC No 06-003 HCSC Yes MH 0: Cured Hepatitis B 06-004 HCSC No 06-005 HCSC No 06-006 HCSC No 06-007 HCSC Yes MH Cerebrovascular Disease 06-009 HCSC No 07-001 HUBA Yes 09-001 HUJF Yes 09-002 HUJF Yes MH Arterial Hypertension BLArterial Hypertension MH Arterial Hypertension MH 0: Atrial Fibrillation 09-003 HUJF Yes MH Depression BL O: Ascites 10-001 HVAL Yes BL Arterial Hypertension Dyslipemia Anxiety BL BL10-002 HVAL Yes MH Arthrosis MH O: Polimialgia Reumatica MH 0: Lichen Planus MH 0: Varicose Veins 10-003 HVAL Yes BL Arterial Hypertension MH Arterial Hy
MH Dyslipemia
MH O: Trombosi 11-001 IVOG Yes Arterial Hypertension 11-002 IVOG Yes 0: Trombosis Venosa Profunda MH 12-001 HUVR No Hypothiroidism 12-002 HUVR Yes MH MH Dyslipemia 12-003 HUVR Yes MH Obesity MH Depression

\_\_\_\_\_\_

<sup>\*0 -</sup> Other

<sup>\*</sup>MH - Medical History, BL - Baseline

Listing 5. Medical History. Relevant Comorbidities. Intention to Treat.

| Time | | | | |
|--------|---------|-------------|-------|--------------------------------|
| Subjid | Site Co | morbidities | point | Туре |
| 12-004 | HUVR | Yes | MH | O: Chronic Renal Disease |
| | | | MH | Depression |
| | | | MH | O: Chronic Leg Ischemya |
| | | | MH | Hypothiroidism |
| | | | MH | O: Chronic Renal Disease |
| 13-001 | HVVA | Yes | MH | Arterial Hypertension |
| 14-001 | HCVA | Yes | MH | Dyslipemia |
| | | | MH | O: Parietotemporal Hematoma Su |
| | | | MH | Depression |
| 15-001 | HUDP | Yes | MH | Arterial Hypertension |
| | | | MH | Dyslipemia |
| 15-002 | HUDP | Yes | MH | Arterial Hypertension |
| | | | MH | Dyslipemia |
| | | | MH | O: Osteoporosis |
| | | | | - |

\_\_\_\_\_

<sup>\*0 -</sup> Other

<sup>\*</sup>MH - Medical History, BL - Baseline

Table 8. Initial Ovarian Cancer Diagnosis History. Descriptive Statistics. Intention to Treat.

| intention to freat. | |
|---|---|
| | Total<br>(n=43) |
| Age at ovarian cancer diagnosis N N Miss Mean Std Dev Median q1 q3 Minimum Maximum | 43<br>0 ( 0.0%)<br>71.4<br>4.5<br>71.0<br>69.0<br>74.0<br>62 |
| Age<br>Missing<br>Less than 70 Years<br>70-80 Years<br>More than 80 Years | 0 ( 0.0%)<br>12 ( 27.9%)<br>29 ( 67.4%)<br>2 ( 4.7%) |
| Weight N N Miss Mean Std Dev Median q1 q3 Minimum Maximum | 32<br>11 ( 25.6%)<br>65.1<br>10.9<br>64.5<br>56.5<br>72.0<br>42 |
| Weight Missing Less than 70Kg 70 - 75 Kg 75 - 80 Kg More than 80Kg | 11 ( 25.6%)<br>21 ( 48.8%)<br>6 ( 14.0%)<br>2 ( 4.7%)<br>3 ( 7.0%) |
| ECOG Missing 0 1 2 3 4 Unknown | 8 ( 18.6%) 14 ( 32.6%) 8 ( 18.6%) 4 ( 9.3%) 0 ( 0.0%) 0 ( 0.0%) 9 ( 20.9%) |

Table 8. Initial Ovarian Cancer Diagnosis History. Descriptive Statistics. Intention to Treat.

| | Total |
|---------------------------------------------|--------------|
| | (n=43) |
| Existence of measurable disease | |
| Missing | 1 ( 2.3%) |
| Yes | 35 ( 81.4%) |
| No | 7 ( 16.3%) |
| Existence of huller discours | |
| Existence of bulky disease Missing | 1 ( 2.3%) |
| Yes | 23 ( 53.5%) |
| No | 19 ( 44.2%) |
| NO | 19 ( 44.2//) |
| Tumor histology | |
| Missing | 1 ( 2.3%) |
| | 40 ( 93.0%) |
| High grade fallopian tube cancer | 1 ( 2.3%) |
| High grade primary peritoneal cancer | 1 ( 2.3%) |
| FIGO Stage | |
| Missing | 3 ( 7.0%) |
| IA | 2 ( 4.7%) |
| IB | 0 ( 0.0%) |
| IC1 | 1 ( 2.3%) |
| IC2 | 0 ( 0.0%) |
| IC3 | 0 ( 0.0%) |
| IIA | 0 ( 0.0%) |
| IIB | 0 ( 0.0%) |
| IIIA1 | 2 ( 4.7%) |
| IIIA2 | 1 ( 2.3%) |
| IIIB | 3 ( 7.0%) |
| IIIC | 22 ( 51.2%) |
| IVA | 0 ( 0.0%) |
| IVB | 5 ( 11.6%) |
| Unknown | 4 ( 9.3%) |
| Other (Specify) | 0 ( 0.0%) |
| Brain metastasis | |
| Missing | 0 ( 0.0%) |
| Yes | 0 ( 0.0%) |
| No | 43 (100.0%) |
| Homologous recombination genes deficiencies | |
| No | 42 ( 97.7%) |
| Yes | 1 ( 2.3%) |
| | 1 ( 2.5%) |

Table 8. Initial Ovarian Cancer Diagnosis History. Descriptive Statistics. Intention to Treat.

| | Total |
|---------------------------------------------|-------------|
| | (n=43) |
| Existence of measurable disease | |
| Missing | 1 ( 2.3%) |
| Yes | 35 ( 81.4%) |
| No | 7 ( 16.3%) |
| Existence of bulky disease | |
| Missing | 1 ( 2.3%) |
| Yes | 23 ( 53.5%) |
| No | 19 ( 44.2%) |
| Tumor histology | |
| Missing | 1 ( 2.3%) |
| High grade serous ovarian cancer | 40 ( 93.0%) |
| High grade fallopian tube cancer | 1 ( 2.3%) |
| High grade primary peritoneal cancer | 1 ( 2.3%) |
| | - ( |
| FIGO Stage | |
| Missing | 3 ( 7.0%) |
| IA | 2 ( 4.7%) |
| IB | 0 ( 0.0%) |
| IC1 | 1 ( 2.3%) |
| IC2 | 0 ( 0.0%) |
| IC3 | 0 ( 0.0%) |
| IIA | 0 ( 0.0%) |
| IIB | 0 ( 0.0%) |
| IIIA1 | 2 ( 4.7%) |
| IIIA2 | 1 ( 2.3%) |
| IIIB | 3 ( 7.0%) |
| IIIC | 22 ( 51.2%) |
| IVA | 0 ( 0.0%) |
| IVB | 5 ( 11.6%) |
| Unknown | 4 ( 9.3%) |
| Other (Specify) | 0 ( 0.0%) |
| Brain metastasis | |
| Missing | 0 ( 0.0%) |
| Yes | 0 ( 0.0%) |
| No | 43 (100.0%) |
| Homologous recombination genes deficiencies | |
| No | 42 ( 97.7%) |
| Yes | 1 ( 2.3%) |

Table 9. Laboratory Initial Ovarian Cancer Diagnosis. Descriptive Statistics. Intention to Treat.

| | Total |
|---------------------------------|-------------|
| | (n=43) |
| Absolute Neutrophils (cells/nL) | |
| N | 36 |
| N Miss | 7 ( 16.3%) |
| Mean | 4853.9 |
| Std Dev | 2210.2 |
| Median | 4610.0 |
| q1 | 3175.0 |
| q3 | 6075.0 |
| Minimum | 1300 |
| Maximum | 11E3 |
| Absolute Neutrophils (cells/nL) | |
| Missing | 7 ( 16.3%) |
| Less than 1500 | 1 ( 2.3%) |
| 1500-8000 | 31 ( 72.1%) |
| More than 8000 | 4 ( 9.3%) |
| Hemoglobin (g/dL) | |
| N | 37 |
| N Miss | 6 ( 14.0%) |
| Mean | 12.0 |
| Std Dev | 1.3 |
| Median | 12.1 |
| q1 | 11.1 |
| q3 | 12.7 |
| Minimum | 9 |
| Maximum | 15 |
| Hemoglobin (g/dL) | |
| Missing | 6 ( 14.0%) |
| Less than 11.6 | 12 ( 27.9%) |
| 11.6-15.0 | 24 ( 55.8%) |
| More than 15.0 | 1 ( 2.3%) |

Table 9. Laboratory Initial Ovarian Cancer Diagnosis. Descriptive Statistics. Intention to Treat.

| | Total |
|----------------------------------|------------------|
| | (n=43) |
| CA125 (U/mL) | |
| N | 35 |
| N Miss | 8 ( 18.6%) |
| Mean | 959.0 |
| Std Dev | 1228.2 |
| Median | 469.8 |
| q1 | 185.6 |
| q3 | 1242.7 |
| Minimum | 8 |
| Maximum | 5879 |
| CA125 (U/mL) | |
| Missing | 8 ( 18.6%) |
| Less than 46.0 | 4 ( 9.3%) |
| 46.0-200.0 | 6 ( 14.0%) |
| 46.0-1000.0 | 15 ( 34.9%) |
| More than 1000.0 | 10 ( 23.3%) |
| Deficiencis in other genes | |
| Missing | 0 ( 0.0%) |
| Yes | 1 ( 2.3%) |
| No | 42 ( 97.7%) |
| Variant classification | |
| Missing | 1 ( 2.3%) |
| Pathogenic | 3 ( 7.0%) |
| Probably pathogenic | 0 ( 0.0%) |
| Variant of uncertain significant | (VOUS) 2 ( 4.7%) |
| Unknown | 37 ( 86.0%) |

Listing 6. Initial Ovarian Cancer Diagnosis History. Intention to Treat.

| Subjid | | _ | | OG Me | asurable | Histo | | | | FIGO |
|---|---|---|---|---|---|---|---|---|---|---|
| 01-001 | HU | В | 74 | 1 | Yes | HG | serous | ovarian | cancer | Unknown |
| 01-002 | HU | В | 73 | 1 | No | HG | serous | ovarian | cancer | IIIC |
| 02-001 | HR | YC | 72 | Missing | Yes | HG | primary | y perito | neal cancer | IIIC |
| 02-002 | HR | YC | 81 | _ | Yes | | - | ovarian | | IIIC |
| 03-001 | IC | OG | 62 | 0 | Yes | HG | serous | ovarian | cancer | IA |
| 03-002 | IC | OG | 71 | Unknown | Yes | HG | serous | ovarian | cancer | IIIC |
| 04-001 | HL | ΕO | 75 | Unknown | Yes | HG | serous | ovarian | cancer | Missing |
| 04-002 | HL | ΕO | 71 | Unknown | Yes | HG | serous | ovarian | cancer | IIIB |
| 04-003 | HL | ΕO | 71 | Missing | Yes | HG | serous | ovarian | cancer | IIIC |
| 04-004 | HL | ΕO | 72 | Unknown | Yes | HG | serous | ovarian | cancer | IC1 |
| 04-005 | HL | ΕO | 71 | Missing | No | HG | serous | ovarian | cancer | Unknown |
| 04-006 | HL | ΕO | 85 | Missing | Missing | HG | serous | ovarian | cancer | Missing |
| 04-007 | HL | ΕO | 75 | 2 | Yes | HG | serous | ovarian | cancer | Missing |
| 04-008 | HL | ΕO | 70 | Missing | Yes | HG | serous | ovarian | cancer | IIIB |
| 05-002 | HU | RS | 77 | Missing | Yes | HG | serous | ovarian | cancer | IIIC |
| 05-003 | HU | RS | 70 | Unknown | Yes | HG | serous | ovarian | cancer | IIIC |
| 05-004 | HU | RS | 71 | Unknown | Yes | HG | serous | ovarian | cancer | Unknown |
| 05-006 | HU | RS | 68 | Missing | Yes | HG | serous | ovarian | cancer | Unknown |
| 06-001 | HC | SC | 74 | 0 | Yes | HG | serous | ovarian | cancer | IVB |
| 06-002 | HC | SC | 69 | 0 | Yes | HG | serous | ovarian | cancer | IIIA1 |
| 06-003 | HC | SC | 67 | 0 | Yes | HG | fallop | ian tube | cancer | IIIC |
| 06-004 | HC | SC | 65 | 0 | Yes | HG | serous | ovarian | cancer | IIIC |
| 06-005 | HC | SC | 66 | Unknown | Yes | HG | serous | ovarian | cancer | IIIC |
| 06-006 | HC | SC | 67 | 0 | Yes | HG | serous | ovarian | cancer | IIIC |
| 06-007 | HC | SC | 79 | Missing | Yes | HG | serous | ovarian | cancer | IVB |
| 06-009 | HC | SC | 73 | 1 | No | HG | serous | ovarian | cancer | IIIC |
| 07-001 | HU: | BA | 71 | 0 | Yes | HG | serous | ovarian | cancer | IVB |
| 09-001 | HU | JF | 72 | 0 | Yes | HG | serous | ovarian | cancer | IIIC |
| 09-002 | HU | JF | 74 | 1 | Yes | HG | serous | ovarian | cancer | IIIC |
| 09-003 | HU | JF | 74 | 0 | Yes | HG | serous | ovarian | cancer | IIIA2 |
| 10-001 | HV. | AL | 71 | 2 | Yes | HG | serous | ovarian | cancer | IIIC |
| 10-002 | HV. | AL | 76 | 2 | Yes | HG | serous | ovarian | cancer | IIIC |
| 10-003 | | | 62 | 0 | No | HG | serous | ovarian | cancer | IA |
| 11-001 | | | 65 | | No | | | ovarian | cancer | |
| 11-002 | IV | OG | 66 | 0 | No | Mi | ssing | | | IIIA1 |
| 12-001 | HU' | VR. | 70 | Unknown | Yes | HG | serous | ovarian | cancer | IVB |
| 12-002 | HU | VR | 70 | 0 | Yes | HG | serous | ovarian | cancer | IIIC |
| 12-003 | | | 69 | 2 | Yes | HG | serous | ovarian | cancer | IIIC |
| 12-004 | HU | VR. | 75 | 1 | Yes | HG | serous | ovarian | cancer | IIIC |
| 13-001 | HV | VA | 69 | 1 | Yes | HG | serous | ovarian | cancer | IIIB |
| 14-001 | HC. | VA<br> | 73 | Unknown | No | HG | serous | ovarian | cancer | IIIC |

\*MG - High Grade

Listing 6. Initial Ovarian Cancer Diagnosis History. Intention to Treat.

| Subjid | Site | Age | EC | OG | Measurable | Histo: | logy | | <br>FIGO |
|---|---|---|---|---|---|---|---|---|---|
| 15-001<br>15-002 | | DP<br>DP | | _ | Yes<br>Yes | | | ovarian<br>ovarian | <br>INB |

\*MG - High Grade

Table 10. Ovarian Cancer Treatments. Previous Surgery. Descriptive Statistics. Intention to Treat.

| | Total<br>(n=43) |
|---------------------------------|-----------------|
| <br>Surgeries | |
| N N | 38 |
| N Miss | 5 ( 11.6%) |
| Mean | 1.2 |
| Std Dev | 0.4 |
| Median | 1.0 |
| q1 | 1.0 |
| q3 | 1.0 |
| Minimum | 1 |
| Maximum | 2 |
| Number of Surgeries per Patient | |
| 0 | 5 ( 11.6%) |
| 1 | 29 ( 67.4%) |
| 2 | 9 ( 20.9%) |
| more than 3 | 0 ( 0.0%) |
| When was surgery performed? | |
| Before relapse (primary) | 41 ( 87.2%) |
| At relapse | 6 ( 12.8%) |
| Surgery type | |
| Missing | 2 ( 4.3%) |
| Primary Debulking Surgery | 23 ( 48.9%) |
| Interval Debulking Surgery | 15 ( 31.9%) |
| Secondary Cytoreduction | 7 ( 14.9%) |
| Surgery outcome | |
| Missing | 1 ( 2.1%) |
| RO | 20 ( 42.6%) |
| R>0 | 10 ( 21.3%) |
| Unknown | 16 ( 34.0%) |

Table 11. Ovarian Cancer. Previous Systemic Treatments.

| | Total<br>(n=43) |
|------------------------------------------|-----------------|
| N. of Prev. Treatments Lines per Patient | |
| N | 43 |
| N Miss | 0 ( 0.0%) |
| Mean | 2.6 |
| Std Dev | 1.3 |
| Median | 2.0 |
| q1 | 2.0 |
| q3 | 4.0 |
| Minimum | 1 |
| Maximum | 6 |
| Prev. Treatments Lines per Patient | |
| 0 | 0 ( 0.0%) |
| 1 or 2 Lines | 25 ( 58.1%) |
| 3 or 4 Lines | 15 ( 34.9%) |
| 5 or more Lines | 3 ( 7.0%) |
| Setting | |
| Before relapse | 71 ( 64.0%) |
| At relapse | 40 ( 36.0%) |
| Line | |
| Maintenance | 23 ( 20.7%) |
| First | 43 ( 38.7%) |
| Second | 28 ( 25.2%) |
| Third | 12 ( 10.8%) |
| Fourth | 4 ( 3.6%) |
| Fifth | 1 ( 0.9%) |
| Sixth | 0 ( 0.0%) |
| Seventh | 0 ( 0.0%) |
| Eighth | 0 ( 0.0%) |
| Ninth | 0 ( 0.0%) |
| Tenth | 0 ( 0.0%) |

<sup>\*(</sup>CL) - Clinical Trial

Table 11. Ovarian Cancer. Previous Systemic Treatments.

| | Total |
|-----------------------------------------------|-------------|
| | (n=43) |
| Treatment type | |
| Amg386 (Trinova Trial) | 1 ( 0.9%) |
| Atezolizumab-Niraparib-Cobimetinib (CT) | 1 ( 0.9%) |
| Bevacizumab | 16 ( 14.4%) |
| Carboplatin | 2 ( 1.8%) |
| Carboplatin-Bevacizumab-Paclitaxel | 6 ( 5.4%) |
| Carboplatin-Caelyx | 14 ( 12.6%) |
| Carboplatin-Gemcitabine | 9 ( 8.1%) |
| Carboplatin-Gemcitabine-Bevacizumab | 3 ( 2.7%) |
| Carboplatin-Paclitaxel | 47 ( 42.3%) |
| Carboplatin-Paclitaxel-Veliparib/Placebo (CT) | 1 ( 0.9%) |
| Docetaxel-Ciclofosfamide | 1 ( 0.9%) |
| Farletuzumab-Pld-Carboplatin | 1 ( 0.9%) |
| Gexmab 25201 (CT) | 1 ( 0.9%) |
| Niraparib | 2 ( 1.8%) |
| Olaparib | 2 ( 1.8%) |
| Pankomab (CT) | 1 ( 0.9%) |
| Pembrolizumab (CT) | 2 ( 1.8%) |
| Rucaparib/Placebo (Ariel Trial) | 1 ( 0.9%) |
| Reason end of treatment | |
| Toxicity | 10 ( 9.0%) |
| Doctor's decision | 9 ( 8.1%) |
| Patient's decision | 1 ( 0.9%) |
| Progression | 28 ( 25.2%) |
| Treatment completed | 59 ( 53.2%) |
| Medium Cytoreductive Laparotomy | 1 ( 0.9%) |
| Microondas Hepatic | 1 ( 0.9%) |
| Unknown | 2 ( 1.8%) |
| Best Radiological Response (RECIST) | |
| Complete Response (CR) | 34 ( 30.6%) |
| Partial Response (PR) | 32 ( 28.8%) |
| Stable Disease (SD) | 32 ( 28.8%) |
| Progressive Disease (PD) | 6 ( 5.4%) |
| Not assessable | 7 ( 6.3%) |
| Treatment free interval | |
| <6 months | 39 ( 35.1%) |
| 6-12 months | 38 ( 34.2%) |
| >12 months | 34 ( 30.6%) |

<sup>\*(</sup>CL) - Clinical Trial

Table 11. Ovarian Cancer. Previous Systemic Treatments.

| | Total<br>(n=43) |
|----------------------------------------|-----------------|
| Previous Platin treatment | |
| Yes | 56 ( 50.5%) |
| No | 6 ( 5.4%) |
| Not applicable (no previous treatment) | 49 ( 44.1%) |

\*(CL) - Clinical Trial

Table 12. Ovarian Cancer. Subsequent Treatments.

| | Total<br>(n=43) |
|------------------------------------------|-----------------|
| W. of Post. Treatments Lines per Patient | |
| N | 32 |
| N Miss | 11 ( 25.6%) |
| Mean | 2.4 |
| Std Dev | 1.2 |
| Median | 2.0 |
| q1 | 1.0 |
| q3 | 3.0 |
| Minimum | 1 |
| Maximum | 5 |
| Post. Treatments Lines per Patient | |
| 0 Lines | 11 ( 25.6%) |
| 1 or 2 Lines | 17 ( 39.5%) |
| 3 or 4 Lines | 13 ( 30.2%) |
| 5 or more Lines | 2 ( 4.7%) |
| Best response | |
| Complete Response (CR) | 1 ( 1.4%) |
| Partial Response (PR) | 21 ( 28.4%) |
| Stable Disease (SD) | 27 ( 36.5%) |
| Progression (PD) | 14 ( 18.9%) |
| Progressive Disease (PD) | 0 ( 0.0%) |
| Not assessable | 11 ( 14.9%) |

Table 12. Ovarian Cancer. Subsequent Treatments.

| | Total |
|--------------------------------------------------------|-------------|
| | (n=43) |
| Drug/Combination name | |
| Bevacizumab | 1 ( 1.3%) |
| Bevacizumab-Cyclophosphamide | 5 ( 6.5%) |
| Bevacizumab-cyclophosphamide<br>Bevacizumab-Paclitaxel | 1 ( 1.3%) |
| | 1 ( 1.3%) |
| Bevacizumab-Topotecan | 4 ( 5.2%) |
| Carboplatin | 2 ( 2.6%) |
| Carboplatin-Bevacizumab-Gembcitabine | |
| Carboplatin-DLP | 4 ( 5.2%) |
| Carboplatin-Gemcitabine | 9 ( 11.7%) |
| Carboplatin-Paclitaxel | 12 ( 15.6%) |
| Carboplatin-Taxol | 1 ( 1.3%) |
| Cisplatin | 2 ( 2.6%) |
| Cisplatin-Gemcitabine | 4 ( 5.2%) |
| Cyclophosfamide | 1 ( 1.3%) |
| DLP | 3 ( 3.9%) |
| Etoposide | 1 ( 1.3%) |
| Folfox | 1 ( 1.3%) |
| Gemcitabine | 4 ( 5.2%) |
| Genoxal | 1 ( 1.3%) |
| Niraparib | 3 ( 3.9%) |
| Olaparib | 7 ( 9.1%) |
| Oxaliplatin | 1 ( 1.3%) |
| Oxaliplatin-Gemcitabine | 1 ( 1.3%) |
| Paclitaxel | 5 ( 6.5%) |
| Topotecan | 2 ( 2.6%) |
| Vb111-Paclitaxel (CT) | 1 ( 1.3%) |
| Reason end of treatment | |
| Progression | 33 ( 44.6%) |
| Toxicity | 15 ( 20.3%) |
| Doctor's decision | 17 ( 23.0%) |
| Patient's decision | 1 ( 1.4%) |
| Death | 1 ( 1.4%) |
| Completed | 2 ( 2.7%) |
| Other | 4 ( 5.4%) |
| Unknown | 1 ( 1.4%) |
| Ongoing? | |
| Ongoing? | 74 ( 06 45) |
| No<br>V | 74 ( 96.1%) |
| Yes | 3 ( 3.9%) |

#### 10.3 Outcome data

### PFS for trabectedin+PLD treatment (43 patients):

Figure 1. Progression Free Survival. Kaplan-Meier Estimates. Per Protocol.



Median PFS = 7.7 months. IC 95: (4.4, 9.4)

## PFS for platin-containing regimens when given right after trabectedin+PLD (27 patients):



# PFS listings for trabectedin+PLD treatment:

Listing 7. Progression Free Survival. Full Analysis Set.

| Subjid Site Start Date PFS Date PFS Event* | Subiid | Site | Start Date | DES Data | DES Fronts | |
|---|---|---|---|---|---|---|
| 04-007 HLEO 04-JUL-2016 15-JUL-2016 0.36 1 02-001 HRYC 08-SEP-2016 06-DCT-2016 0.92 1 04-006 HLEO 09-DCT-2017 19-NOV-2017 1.35 1 15-002 HUDP 27-MAY-2016 18-JUL-2016 1.71 1 12-004 HUVR 12-DEC-2017 06-FEB-2018 1.84 1 09-003 HUJF 23-MAY-2019 24-JUL-2019 2.04 1 15-001 HUDP 15-FEB-2016 23-APR-2016 2.23 1 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-DCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 7.56 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-003 HUSS 22-MAR-2017 29-NOV-2017 8.28 1 06-009 HCSC 12-FEB-2018 11-DCT-2018 7.92 0 05-003 HURS 22-MAR-2017 05-FEB-2018 8.41 1 04-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HCSC 07-AUG-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 15-FEB-2018 8.41 1 04-001 HCSC 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2017 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCSO 29-NOV-2017 17-SEP-2018 9.60 1 14-001 HCSO 29-NOV-2017 18-JAN-2018 9.69 1 10-002 HUB 27-MAR-2015 16-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 12-Z048 9.69 1 10-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 | | | | | | |
| 04-007 HLEO 04-JUL-2016 15-JUL-2016 0.36 1 02-001 HRYC 08-SEP-2016 06-DCT-2016 0.92 1 04-006 HLEO 09-DCT-2017 19-NOV-2017 1.35 1 15-002 HUDP 27-MAY-2016 18-JUL-2016 1.71 1 12-004 HUVR 12-DEC-2017 06-FEB-2018 1.84 1 09-003 HUJF 23-MAY-2019 24-JUL-2019 2.04 1 15-001 HUDP 15-FEB-2016 23-APR-2016 2.23 1 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-DCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 7.56 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-003 HUSS 22-MAR-2017 29-NOV-2017 8.28 1 06-009 HCSC 12-FEB-2018 11-DCT-2018 7.92 0 05-003 HURS 22-MAR-2017 05-FEB-2018 8.41 1 04-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HCSC 07-AUG-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 15-FEB-2018 8.41 1 04-001 HCSC 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2017 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCSO 29-NOV-2017 17-SEP-2018 9.60 1 14-001 HCSO 29-NOV-2017 18-JAN-2018 9.69 1 10-002 HUB 27-MAR-2015 16-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2016 12-Z048 9.69 1 10-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 | 06-001 | HC SC | 29-0CT-2019 | 03-NOV-2019 | 0.16 | 1 |
| O2-001 | 10-002 | HVAL | 08-MAY-2015 | 15-MAY-2015 | 0.23 | 1 |
| 04-006 | 04-007 | HLEO | 04-JUL-2016 | 15-JUL-2016 | 0.36 | 1 |
| 04-006 | 02-001 | HRYC | 08-SEP-2016 | 06-0CT-2016 | 0.92 | 1 |
| 12-004 HUVR 12-DEC-2017 06-FEB-2018 1.84 1 09-003 HUJF 23-MAY-2019 24-JUL-2019 2.04 1 15-001 HUDP 15-FEB-2016 23-APR-2016 2.23 1 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-OCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 014-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2019 8.38 1 06-007 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2017 13-MAR-2019 9.40 1 11-001 HVAL 29-MAY-2017 13-MAR-2018 9.46 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.69 1 11-001 HUB 20-MAY-2017 18-JAN-2018 9.69 1 12-003 HUR 29-MAR-2017 18-JAN-2018 9.69 1 12-003 HUR 29-MAR-2017 18-JAN-2018 9.69 1 11-002 HUB 27-MAR-2019 15-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 12-EB-2017 10.12 1 01-002 HUB 27-MAR-2019 12-EB-2017 10.12 1 01-002 HUB 27-MAR-2019 15-FEB-2016 12-22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12-EB 10-001 12-EB-2017 10.12 1 01-002 HUB 27-MAR-2019 15-FEB-2016 12-22 1 01-001 HUB 20-MAY-2016 12-Z2-MAR-2017 13.41 1 | | HLEO | 09-0CT-2017 | 19-NOV-2017 | 1.35 | |
| 09-003 HUJF 23-MAY-2019 24-JUL-2019 2.04 1 15-001 HUDP 15-FEB-2016 23-APR-2016 2.23 1 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-OCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-004 HCSC 07-AUG-20 | | | | | | |
| 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-OCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOY-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-004 HCSC 12-FEB-20 | 12-004 | | | | | 1 |
| 07-001 HUBA 28-AUG-2015 13-NOV-2015 2.53 1 06-002 HCSC 25-OCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOY-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-004 HCSC 12-FEB-20 | 09-003 | HUJF | 23-MAY-2019 | 24-JUL-2019 | 2.04 | 1 |
| 06-002 HCSC 25-OCT-2019 13-JAN-2020 2.63 1 06-005 HCSC 13-FEB-2018 21-MAY-2018 3.19 1 05-004 HURS 07-JAN-2015 06-MAY-2015 3.91 1 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 10-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-004 HVAL 28-JUL-20 | | HUDP | 15-FEB-2016 | 23-APR-2016 | 2.23 | |
| 06-005 | 07-001 | HUBA | 28-AUG-2015 | 13-NOV-2015 | 2.53 | 1 |
| 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-20 | 06-002 | HC SC | 25-OCT-2019 | 13-JAN-2020 | 2.63 | 1 |
| 03-001 ICOG 17-SEP-2019 24-JAN-2020 4.24 1 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-20 | 06-005 | HC SC | 13-FEB-2018 | 21-MAY-2018 | 3.19 | 1 |
| 04-004 HLEO 06-NOV-2017 20-MAR-2018 4.40 1 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-20 | | HURS | 07-JAN-2015 | 06-MAY-2015 | 3.91 | 1 |
| 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-FEB-2018 8.41 1 04-001 HLEO 17-MAY-20 | 03-001 | ICOG | 17-SEP-2019 | 24-JAN-2020 | 4.24 | 1 |
| 04-005 HLEO 04-MAY-2017 19-SEP-2017 4.53 1 12-002 HUVR 18-DEC-2018 16-MAY-2019 4.90 1 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-FEB-2018 8.41 1 04-001 HLEO 17-MAY-20 | 04-004 | HLEO | 06-NOV-2017 | 20-MAR-2018 | 4.40 | 1 |
| 02-002 HRYC 16-NOV-2018 26-APR-2019 5.29 0 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-20 | | HLEO | 04-MAY-2017 | 19-SEP-2017 | 4.53 | |
| 06-006 HCSC 08-MAR-2019 30-AUG-2019 5.75 1 06-003 HCSC 14-SEP-2017 06-APR-2018 6.70 1 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-20 | | | | | | |
| 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 10-002 HUB 27-MAR-201 | | | | | | |
| 06-004 HCSC 07-AUG-2018 28-FEB-2019 6.74 1 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 10-002 HUB 27-MAR-201 | 06-006 | HC SC | 08-MAR-2019 | 30-AUG-2019 | 5.75 | 1 |
| 10-003 HVAL 21-JAN-2019 08-SEP-2019 7.56 1 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 | 06-003 | HC SC | 14-SEP-2017 | 06-APR-2018 | 6.70 | 1 |
| 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 | | | | | | |
| 10-001 HVAL 28-JUL-2015 18-MAR-2016 7.69 1 06-009 HCSC 12-FEB-2018 11-OCT-2018 7.92 0 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 | 10-003 | HVAL | 21-JAN-2019 | 08-SEP-2019 | 7.56 | 1 |
| 05-003 HURS 22-MAR-2017 29-NOV-2017 8.28 1 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO | | HVAL | 28-JUL-2015 | 18-MAR-2016 | 7.69 | |
| 04-002 HLEO 20-JUN-2018 02-MAR-2019 8.38 1 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 06-007 HCSC 25-MAY-2017 05-FEB-2018 8.41 1 04-001 HLEO 17-MAY-2016 02-FEB-2017 8.58 0 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 04-002 | HLEO | 20-JUN-2018 | 02-MAR-2019 | 8.38 | 1 |
| 05-006 HURS 18-MAY-2015 15-FEB-2016 8.97 1 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 06-007 | HC SC | 25-MAY-2017 | 05-FEB-2018 | 8.41 | 1 |
| 11-001 IVOG 15-APR-2015 26-JAN-2016 9.40 1 14-001 HCVA 29-MAY-2017 13-MAR-2018 9.46 1 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 05-006 | | | | | 1 |
| 04-008 HLEO 29-NOV-2017 17-SEP-2018 9.60 1 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 11-001 | IVOG | 15-APR-2015 | 26-JAN-2016 | 9.40 | 1 |
| 12-003 HUVR 29-MAR-2017 18-JAN-2018 9.69 1 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | 1 |
| 09-001 HUJF 11-APR-2016 13-FEB-2017 10.12 1 01-002 HUB 27-MAR-2019 06-FEB-2020 10.38 1 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 12-003 | HUVR | 29-MAR-2017 | 18-JAN-2018 | 9.69 | 1 |
| 11-002 IVOG 19-JAN-2015 26-JAN-2016 12.22 1 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0 04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1 09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | 09-001 | HUJF | 11-APR-2016 | 13-FEB-2017 | 10.12 | 1 |
| 01-001 HUB 20-MAY-2016 15-JUN-2017 12.85 0<br>04-003 HLEO 08-FEB-2016 22-MAR-2017 13.41 1<br>09-002 HUJF 21-OCT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 09-002 HUJF 21-0CT-2015 10-DEC-2016 13.67 1 | | | | | | |
| 09-002 HUJF 21-0CT-2015 10-DEC-2016 13.67 1 | 01-001 | HUB | 20-MAY-2016 | 15-JUN-2017 | 12.85 | 0 |
| | | HLEO | 08-FEB-2016 | 22-MAR-2017 | 13.41 | 1 |
| 03-002 ICOG 15-MAY-2017 07-SEP-2018 15.77 1 | | | | | | |
| | 03-002 | ICOG | 15-MAY-2017 | 07-SEP-2018 | 15.77 | 1 |

\*Events: Progression or death by treatment

Patients censored at post treatment or lost to follow up

Listing 7. Progression Free Survival. Full Analysis Set.

| Subjid | Site | Start Date | PFS Date | PFS Even | t* |
|--------|------|-------------|-------------|----------|----|
| 13-001 | HVVA | 07-MAY-2015 | 20-FEB-2017 | 21.52 | 1 |
| 05-002 | HURS | 09-NOV-2017 | 07-DCT-2019 | 22.91 | 1 |
| 12-001 | HUVR | 25-JUL-2017 | 22-JUN-2021 | 46.93 | 1 |

\*Events: Progression or death by treatment

Patients censored at post treatment or lost to follow up

### Overall survival for trabectedin+PLD treatment:

Figure 2. Overall Survival. Kaplan-Meier Estimates. Full Analysis Set.



 $\label{eq:Median OS = 19.5 months. IC 95: (12.8, 27.2)} \ \ \\$ 

Listing 8. Overall Survival. Full Analysis Set.

| Subjid | Site | Start Date | OS Date Overa | l Survival Event* | - |
|---|---|---|---|---|---|
| 06-001 | | | 03-NOV-2019 | 0.16 | 1 |
| 10-002 | HVAL | 08-MAY-2015 | 29-MAY-2015 | 0.69 | 1 |
| 02-001 | HRYC | 08-SEP-2016 | 28-0CT-2016 | 1.64 | 1 |
| 12-004 | HUVR | 12-DEC-2017 | 27-FEB-2018<br>09-MAY-2016 | 2.53 | 1 |
| 15-001 | HUDP | 15-FEB-2016 | 09-MAY-2016 | 2.76 | 1 |
| 04-006 | HLEO | 09-DCT-2017 | 12-JAN-2018 | 3.12 | 1 |
| 15-002 | HUDP | 27-MAY-2016 | 03-SEP-2016 | 3.25 | 1 |
| 09-003 | HUJF | 23-MAY-2019 | 27-SEP-2019 | 4.17 | 1 |
| 06-002 | HC SC | 25-OCT-2019 | 07-APR-2020 | 5.42 | 1 |
| 05-004 | HURS | 07-JAN-2015 | 09-JUL-2015 | 6.01 | 1 |
| 04-002 | HLEO | 20-JUN-2018 | 21-FEB-2019 | 8.08 | 0 |
| 12-003 | HUVR | 29-MAR-2017 | 16-FEB-2018 | 10.65 | 1 |
| 06-005 | HC SC | 13-FEB-2018 | 11-JAN-2019 | 10.91 | 1 |
| 07-001 | HUBA | 28-AUG-2015 | 27-JUL-2016 | 10.98 | 1 |
| 10-003 | HVAL | 21-JAN-2019 | 26-DEC-2019<br>11-OCT-2020 | 11.14 | 1 |
| 03-001 | ICOG | 17-SEP-2019 | 11-0CT-2020 | 12.82 | 1 |
| 12-002 | HUVR | 18-DEC-2018 | 06-FEB-2020 | 13.64 | 1 |
| 04-004 | HLEO | 06-NOV-2017 | 15-APR-2019 | 17.25 | 1 |
| 04-003 | HLEO | 08-FEB-2016 | 30-JUL-2017 | 17.68 | 1 |
| 04-007 | HLEO | 04-JUL-2016 | 27-DEC-2017 | 17.78 | 1 |
| 06-003 | HC SC | 14-SEP-2017 | 19-MAR-2019 | 18.11 | 1 |
| 01-002 | HUB | 27-MAR-2019 | 03-NOV-2020 | 19.29 | 1 |
| 10-001 | HVAI. | 28-JUL-2015 | 11-MAR-2017 | 19.45 | 1 |
| 13-001 | HVVA | 07-MAY-2015 | 23-JAN-2017 | 20.60 | 0 |
| 06-004 | HC SC | 07-AUG-2018 | 29-APR-2020 | 20.74 | 1 |
| 04-001 | HLEO | 17-MAY-2016 | 05-MAR-2018 | 21.59 | 1 |
| 01-001 | HUB | 20-MAY-2016 | 10-MAY-2018 | 23.66 | 1 |
| 06-007 | HC SC | 25-MAY-2017 | 21-JUN-2019 | 24.88 | 1 |
| 09-001 | HUJF | 11-APR-2016 | 18-JUL-2018 | 27.21 | 1 |
| 06-009 | HC SC | 12-FEB-2018 | 03-0CT-2020 | 31.68 | 1 |
| 11-002 | IVOG | 19-JAN-2015 | 10-SEP-2017 | 31.71 | 1 |
| 09-002 | HUJF | 21-0CT-2015 | 16-AUG-2018 | 33.85 | 1 |
| 11-001 | IVOG | 15-APR-2015 | 10-APR-2018 | 35.85 | 0 |
| 04-005 | HLEO | 04-MAY-2017 | 26-MAY-2020 | 36.74 | 1 |
| 06-006 | HC SC | 08-MAR-2019 | 22-JUN-2022 | 39.50 | 0 |
| 02-002 | HRYC | 16-NOV-2018 | 08-APR-2022 | 40.72 | 1 |
| 05-002 | HURS | 09-NOV-2017 | 26-0CT-2021 | 47.55 | 0 |
| 04-008 | HLEO | 29-NOV-2017 | 21_FEB_2022 | 50.77 | 0 |
| | | 29-MAY-2017 | | 53.50 | 0 |
| 12-001 | HUVR | 25-JUL-2017 | 21-JAN-2022 | 53.93 | 0 |

-----

\*Events: Death

Patients censored at lost to follow up

Listing 8. Overall Survival. Full Analysis Set.

| Subjid | Site | Start Date | OS Date Ov | eral Survival | Event* |
|---|---|---|---|---|---|
| 03-002<br>05-003<br>05-006 | ICOG<br>HURS<br>HURS | 22-MAR-2017 | 20-DEC-2021<br>15-NOV-2021<br>29-OCT-2020 | 55.2<br>55.8<br>65.4 | 33 0 |

\*Events: Death

Patients censored at lost to follow up

Table 13. Objective Response Rate. Descriptive and Inferential Statistics. Full Analysis Set.

| | Total |
|------------------------------------|-------------|
| | (n=43) |
| Radiological best overall responce | |
| Progression Disease (PD) | 5 ( 11.6%) |
| Stable Disease (SD) | 13 ( 30.2%) |
| Partial Response (PR) | 14 ( 32.6%) |
| Complete Response (CR) | 4 ( 9.3%) |
| Not assessable | 7 ( 16.3%) |
| Biological best overall responce | |
| Progression | 3 ( 7.0%) |
| Stabilization | 3 ( 7.0%) |
| Response | 14 ( 32.6%) |
| Response and normalization | 11 ( 25.6%) |
| Not assessable | 12 ( 27.9%) |
| Objective Response Rate | |
| PD or SD | 18 ( 41.9%) |
| PR or CR | 18 ( 41.9%) |
| NE | 7 ( 16.3%) |

ORR Binomial's confidence interval 95 with 36 patients prob = 0.5 with CI (0.345 - 0.655)
Listing 9. Objective Response Rate. Full Analysis Set.

| Subjid Site Best Response 01-001 HUB Stable Disease (SD) 01-002 HUB Partial Response (PR) 02-001 HRYC Stable Disease (SD) 02-002 HRYC Partial Response (PR) | 21-SEP-2016<br>16-JUN-2019<br>11-OCT-2016<br>19-FEB-2019<br>18-NOV-2019<br>12-JUL-2017 |
|---|---|
| 01-002 HUB Partial Response (PR)<br>02-001 HRYC Stable Disease (SD)<br>02-002 HRYC Partial Response (PR) | 16-JUN-2019<br>11-OCT-2016<br>19-FEB-2019<br>18-NOV-2019<br>12-JUL-2017 |
| 02-001 HRYC Stable Disease (SD)<br>02-002 HRYC Partial Response (PR) | 11-0CT-2016<br>19-FEB-2019<br>18-NOV-2019<br>12-JUL-2017 |
| 02-002 HRYC Partial Response (PR) | 19-FEB-2019<br>18-NOV-2019<br>12-JUL-2017 |
| • | 18-NOV-2019<br>12-JUL-2017 |
| | 12-JUL-2017 |
| 03-001 ICOG Partial Response (PR) | |
| 03-002 ICOG Partial Response (PR) | 12-JUL-2016 |
| 04-001 HLEO Partial Response (PR) | |
| 04-002 HLEO Partial Response (PR) | 05-DEC-2019 |
| 04-003 HLEO Not assessable | |
| 04-004 HLEO Stable Disease (SD) | 14-DEC-2017 |
| 04-005 HLEO Stable Disease (SD) | 19-MAY-2017 |
| 04-006 HLEO Not assessable | |
| 04-007 HLEO Progression Disease (PD) | 15-JUL-2016 |
| 04-008 HLEO Partial Response (PR) | 03-APR-2018 |
| 05-002 HURS Complete Response (CR) | 28-MAY-2018 |
| 05-003 HURS Partial Response (PR) | 06-SEP-2017 |
| 05-004 HURS Stable Disease (SD) | 10-MAR-2015 |
| 05-006 HURS Complete Response (CR) | 21-0CT-2015 |
| 06-001 HCSC Not assessable | |
| 06-002 HCSC Not assessable | |
| 06-003 HCSC Partial Response (PR) | 28-DEC-2017 |
| 06-004 HCSC Stable Disease (SD) | 16-NOV-2018 |
| 06-005 HCSC Progression Disease (PD) | 21-MAY-2018 |
| 06-006 HCSC Partial Response (PR) | 14-JUN-2019 |
| 06-007 HCSC Stable Disease (SD) | 07-NOV-2017 |
| 06-009 HCSC Stable Disease (SD) | 23-APR-2018 |
| 07-001 HUBA Progression Disease (PD) | 13-NOV-2015 |
| 09-001 HUJF Stable Disease (SD) | 26-JUL-2017 |
| 09-002 HUJF Complete Response (CR) | 07-JUL-2016 |
| 09-003 HUJF Not assessable | |
| 10-001 HVAL Partial Response (PR) | 26-0CT-2015 |
| 10-002 HVAL Not assessable | |
| 10-003 HVAL Stable Disease (SD) | 25-APR-2019 |
| 11-001 IVOG Partial Response (PR) | 02-SEP-2015 |
| 11-002 IVOG Complete Response (CR) | 03-JUN-2015 |
| 12-001 HUVR Stable Disease (SD) | 22-SEP-2017 |
| 12-002 HUVR Partial Response (PR) | 05-MAR-2019 |
| 12-003 HUVR Partial Response (PR) | 31-JUL-2017 |
| 12-004 HUVR Not assessable | |
| 13-001 HVVA Stable Disease (SD) | 17-SEP-2015 |

Listing 9. Objective Response Rate. Full Analysis Set.

| Subjid | Site | Best Response | OS Date |
|--------|------|---------------------|------------------|
| 14-001 | HCVA | Stable Disease (SD) | 28-AUG-2017 |
| 15-001 | HUDP | Progression Disease | (PD) 23-APR-2016 |
| 15-002 | HUDP | Progression Disease | (PD) 18-JUL-2016 |

Table 14. Disease Control Rate. Descriptive and Inferential Statistics. Full Analysis Set.

| | Total |
|------------------------------------|-------------|
| | (n=43) |
| Radiological best overall responce | |
| Progression Disease (PD) | 5 ( 11.6%) |
| Stable Disease (SD) | 13 ( 30.2%) |
| Partial Response (PR) | 14 ( 32.6%) |
| Complete Response (CR) | 4 ( 9.3%) |
| Not assessable | 7 ( 16.3%) |
| Biological best overall responce | |
| Progression | 3 ( 7.0%) |
| Stabilization | 3 ( 7.0%) |
| Response | 14 ( 32.6%) |
| Response and normalization | 11 ( 25.6%) |
| Not assessable | 12 ( 27.9%) |
| Objective Response Rate | |
| PD | 5 ( 11.6%) |
| CR or PR or SD | 31 ( 72.1%) |
| NE | 7 ( 16.3%) |

DCR Binomial's confidence interval 95 with 36 patients prob = 0.8611111111 with CI (0.713 - 0.939)

Listing 11. Duration of Response Treatment. Full Analysis Set.

| Response<br>Subjid | _ | sion Progression<br>Best Response | Data tu | | Date Dur | |
|---|---|---|---|---|---|---|
| 545]14 | 2166 | best response | Date ty | pe* | Date Dur | at 1 OH |
| 01-001 | HUB | Stable Disease (SD) | 21-SEP-2016 | | | 0.00 |
| 01-002 | HUB | Partial Response (PR) | 16-JUN-2019 | R | 06-FEB-2020 | 7.72 |
| 02-001 | HRYC | Stable Disease (SD) | 11-0CT-2016 | C | 06-DCT-2016 | 0.00 |
| 02-002 | HRYC | Partial Response (PR) | 19-FEB-2019 | | | 0.00 |
| 03-001 | ICOG | Partial Response (PR) | 18-NOV-2019 | R | 24-JAN-2020 | 2.20 |
| 03-002 | ICOG | Partial Response (PR) | 12-JUL-2017 | R, B (ca 125) | 07-SEP-2018 | 13.87 |
| 04-001 | HLEO | Partial Response (PR) | 12-JUL-2016 | B (ca 125) | 04-FEB-2017 | 6.80 |
| 04-002 | HLEO | Partial Response (PR) | 05-DEC-2019 | R | 02-MAR-2019 | 0.00 |
| 04-003 | HLEO | Not assessable | | R | 22-MAR-2017 | 0.00 |
| 04-004 | HLEO | Stable Disease (SD) | 14-DEC-2017 | R | 20-MAR-2018 | 3.15 |
| 04-005 | HLEO | Stable Disease (SD) | 19-MAY-2017 | R | 19-SEP-2017 | 4.04 |
| 04-006 | HLEO | Not assessable | | R, C, B (ca125) | 19-NOV-2017 | 0.00 |
| 04-007 | HLEO | Progression Disease (PD) | 15-JUL-2016 | R | 15-JUL-2016 | 0.00 |
| 04-008 | HLEO | Partial Response (PR) | 03-APR-2018 | R, B (ca 125) | 17-SEP-2018 | 5.49 |
| 05-002 | HURS | Complete Response (CR) | 28-MAY-2018 | R | 07-DCT-2019 | 16.33 |
| 05-003 | HURS | Partial Response (PR) | 06-SEP-2017 | R | 29-NOV-2017 | 2.76 |
| 05-004 | HURS | Stable Disease (SD) | 10-MAR-2015 | R | 06-MAY-2015 | 1.87 |
| 05-006 | HURS | Complete Response (CR) | 21-0CT-2015 | R | 15-FEB-2016 | 3.84 |
| 06-001 | HC SC | Not assessable | , | C | 03-NOV-2019 | 0.00 |
| 06-002 | HC SC | Not assessable | | R, C | 13-JAN-2020 | 0.00 |
| 06-003 | HC SC | Partial Response (PR) | 28-DEC-2017 | R | 06-APR-2018 | 3.25 |
| 06-004 | HC SC | Stable Disease (SD) | | R | 28-FEB-2019 | 3.42 |
| 06-005 | HC SC | Progression Disease (PD) | 21-MAY-2018 | R, C, B (ca125) | 21-MAY-2018 | 0.00 |
| 06-006 | HC SC | Partial Response (PR) | 14-JUN-2019 | R, B (ca 125) | 30-AUG-2019 | 2.53 |

Duration in months.

Listing 11. Duration of Response Treatment. Full Analysis Set.

| Response | Progress | sion Progression | | | | |
|---|---|---|---|---|---|---|
| Subjid | Site | Best Response | Date ty | pe* | Date Dur | ation |
| 06-007 | HC SC | Stable Disease (SD) | 07-NOV-2017 | R, B (ca 125) | 05-FEB-2018 | 2.96 |
| 06-009 | HC SC | Stable Disease (SD) | 23-APR-2018 | C | 03-NOV-2018 | 6.38 |
| 07-001 | HUBA | Progression Disease (PD) | 13-NOV-2015 | R | 13-NOV-2015 | 0.00 |
| 09-001 | HUJF | Stable Disease (SD) | 26-JUL-2017 | R | 13-FEB-2017 | 0.00 |
| 09-002 | HUJF | Complete Response (CR) | 07-JUL-2016 | R | 10-DEC-2016 | 5.13 |
| 09-003 | HUJF | Not assessable | | C | 24-JUL-2019 | 0.00 |
| 10-001 | HVAL | Partial Response (PR) | 26-0CT-2015 | R, B (ca 125) | 18-MAR-2016 | 4.73 |
| 10-002 | HVAL | Not assessable | | C | 15-MAY-2015 | 0.00 |
| 10-003 | HVAL | Stable Disease (SD) | 25-APR-2019 | C | 08-SEP-2019 | 4.47 |
| 11-001 | IVOG | Partial Response (PR) | 02-SEP-2015 | R, C, B (ca125) | 26-JAN-2016 | 4.80 |
| 11-002 | IVOG | Complete Response (CR) | 03-JUN-2015 | R, C, B (ca125) | 26-JAN-2016 | 7.79 |
| 12-001 | HUVR | Stable Disease (SD) | 22-SEP-2017 | R, B (ca 125) | 22-JUN-2021 | 44.99 |
| 12-002 | HUVR | Partial Response (PR) | 05-MAR-2019 | R, B (ca 125) | 16-MAY-2019 | 2.37 |
| 12-003 | HUVR | Partial Response (PR) | 31-JUL-2017 | R, C | 18-JAN-2018 | 5.62 |
| 12-004 | HUVR | Not assessable | | C | 06-FEB-2018 | 0.00 |
| 13-001 | HVVA | Stable Disease (SD) | 17-SEP-2015 | R | 20-FEB-2017 | 17.15 |
| 14-001 | HCVA | Stable Disease (SD) | 28-AUG-2017 | R | 13-MAR-2018 | 6.47 |
| 15-001 | HUDP | Progression Disease (PD) | 23-APR-2016 | R, C | 23-APR-2016 | 0.00 |
| 15-002 | HUDP | Progression Disease (PD) | 18-JUL-2016 | R, C, B (ca125) | 18-JUL-2016 | 0.00 |

Duration in months.

\_\_\_\_\_\_

<sup>\*</sup>R-Radiological, C-Clinical, B-Biological.

<sup>\*</sup>R-Radiological, C-Clinical, B-Biological.

### 10.4 Main results

Between November 2021 and June 2022, 43 patients were recruited with median age 74 years (70-86). At initial diagnosis, most common FIGO stages were IIIC (51.2%), IVB (11.6%), and IIIB (7.0%). Before trabectedin+PLD (baseline), patients had ECOG performance status 0, 1, or 2 (34.1%, 41.5%, and 9.8%) and 81.4% had measurable disease. The median number of previous lines was 2 (1-6). The initial dose of trabectedin was 1.1 mg/m² in 76.7% of patients (16.3% with <1.1 and 4.7% with >1.1 mg/m²) while 76.7% of patients had PLD at 30 mg (18.6% with <30 mg and 2.3% with >30 mg). The median of trabectedin+PLD cycles was 5 (1-21) and 53.5% of patients had at least one cycle delayed. All patients ended treatment for the following reasons: patient's decision (7.0%), doctor's decision (23.3%), disease progression (39.5%), toxicity (23.83%) and 7.0% due to other factors. Median PFS for the trabectedin+PLD combination was 7.7 months (95% CI 4.4-9.4) with best overall response rates of 4 CR (9.3%), 14 PR (32.6%), 13 SD (30.2%), and 5 PD (11.6%). Median overall survival (OS) was 19.5 months (95% CI 12.8-27.2). Overall, the most common G3-4 hematological events were neutropenia (23.3%), thrombocytopenia (7.0%), and anemia (2.3%), being asthenia (11.6%), mucositis (4.7%), and transaminitis (4.7%) the most frequent G3 nonhematological toxicities.

# 10.5 Other analyses

No other analyses were performed.

10.6 Adverse events/adverse reactions

Table 15.1. Adverse Events by Haematology or Non - Haematology. Descriptive Statistics. Safety Analysis Set.

| _ | | | _ | |
|-----------------------------------|----------|------|---|--------|
| Term | | Tota | | |
| aematological | | | | |
| _ | SUBJECTS | 10 | ( | 23.3%) |
| | EPISODES | 13 | | |
| Neutrophil count decreased | SUBJECTS | 16 | ( | 37.2%) |
| | EPISODES | 26 | | |
| Platelet count decreased | SUBJECTS | 6 | ( | 14.0%) |
| | EPISODES | 6 | | |
| White Blood Cells Decreased | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 4 | | |
| on-Haematological | | | | |
| Abdominal pain | SUBJECTS | 1 | ( | 2.3%) |
| - | EPISODES | 1 | | |
| Alopecia | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Asthenia | SUBJECTS | 21 | ( | 48.8%) |
| | EPISODES | 25 | | |
| Constipation | SUBJECTS | 2 | ( | 4.7%) |
| - | EPISODES | 2 | | |
| Dissociated Cholestasis | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Dysuria | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| General Muscular Pain | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Headache | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Hiporexia | SUBJECTS | 1 | ( | 2.3%) |
| - | EPISODES | 1 | | |
| Hypersensitization To Trabectidin | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Hypertension | SUBJECTS | 2 | ( | 4.7%) |
| | EPISODES | 2 | | |
| Hypokalemia | SUBJECTS | 1 | ( | 2.3%) |
| | EPISODES | 1 | | |
| Mucositis | SUBJECTS | 6 | ( | 14.0%) |
| | EPISODES | 6 | | |
| | SUBJECTS | 10 | ( | 23.3%) |
| Nausea | DODODOLD | | | |
| | EPISODES | 10 | | |
| | EPISODES | | ( | 2.3%) |

Table 15.1. Adverse Events by Haematology or Non - Haematology. Descriptive Statistics. Safety Analysis Set.

\_\_\_\_\_ Haematology Total \_\_\_\_\_ Respiratory Infection SUBJECTS 1 ( 2.3%)
EPISODES 1 SUBJECTS EPISODES SUBJECTS Serum Urea Increased 1 ( 2.3%) 1 Skin Disorders 2 ( 4.7%) EPISODES 2 SUBJECTS 4 ( 9.3%) EPISODES 4 Transaminitis Urinary Tract Infection SUBJECTS 3 ( 7.0%) EPISODES SUBJECTS 6 ( 14.0%) Vomiting EPISODES \_\_\_\_\_\_

Table 15.2. Adverse Events by Grade. Descriptive Statistics. Safety Analysis Set.

\_\_\_\_\_\_ Grade Total \_\_\_\_\_\_ Any grade Abdominal pain SUBJECTS 1 ( 2.3%) EPISODES 1 1 ( 2.3%) Alopecia SUBJECTS EPISODES 1 SUBJECTS 10 ( 23.3%) EPISODES 13 Anemia Asthenia 21 ( 48.8%) SUBJECTS EPISODES 25 SUBJECTS 2 ( 4.7%) Constipation EPISODES SUBJECTS Dissociated Cholestasis 1 ( 2.3%) EPISODES 1 Dysuria SUBJECTS 1 ( 2.3%) EPISODES - 1 1 ( 2.3%) General Muscular Pain SUBJECTS EPISODES 1 Headache SUBJECTS 1 ( 2.3%) EPISODES 1 SUBJECTS Hiporexia 1 ( 2.3%) EPISODES 1 Hypersensitization To Trabectidin SUBJECTS 1 ( 2.3%) EPISODES 1 2 ( 4.7%) Hypertension SUBJECTS EPISODES Hypokalemia SUBJECTS 1 ( 2.3%) EPISODES 1 SUBJECTS Mucositis 6 ( 14.0%) EPISODES Nausea SUBJECTS 10 ( 23.3%) EPISODES 10 16 ( 37.2%) Neutrophil count decreased SUBJECTS EPISODES 26 Palmar-Plantar Erythrodysesthesia SUBJECTS 1 ( 2.3%) 1 EPISODES Platelet count decreased SUBJECTS 6 ( 14.0%) EPISODES 6 Respiratory Infection SUBJECTS 1 ( 2.3%) EPISODES - 1 Serum Urea Increased SUBJECTS 1 ( 2.3%) EPISODES 1

Table 15.2. Adverse Events by Grade. Descriptive Statistics. Safety Analysis Set.

| Grade | | |
|-----------------------------|------------|------------|
| Term | | tal |
| Skin Disorders | SUBJECTS | |
| | EPISODES : | 2 |
| Transaminitis | SUBJECTS | 4 ( 9.3%) |
| | EPISODES 4 | 4 |
| Urinary Tract Infection | SUBJECTS | 3 ( 7.0%) |
| | EPISODES 4 | 4 |
| Vomiting | SUBJECTS | 6 ( 14.0%) |
| | EPISODES | 6 |
| White Blood Cells Decreased | SUBJECTS | 1 ( 2.3%) |
| | EPISODES 4 | 4 |
| Grade 1 | | |
| Abdominal pain | SUBJECTS | 1 ( 2.3%) |
| - | | 1 |
| Alopecia | SUBJECTS | 1 ( 2.3%) |
| • | EPISODES | 1 |
| Anemia | | 4 ( 9.3%) |
| | EPISODES | 7 |
| Asthenia | | 5 ( 11.6%) |
| | | 5 |
| Constipation | | 2 ( 4.7%) |
| • | EPISODES : | 2 |
| Dissociated Cholestasis | | 1 ( 2.3%) |
| | EPISODES | 1 |
| Dysuria | SUBJECTS | 1 ( 2.3%) |
| • | EPISODES | 1 |
| General Muscular Pain | SUBJECTS | 1 ( 2.3%) |
| | EPISODES : | 1 |
| Headache | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Hiporexia | SUBJECTS | 1 ( 2.3%) |
| • | EPISODES | 1 |
| Hypertension | | 2 ( 4.7%) |
| •• | EPISODES : | 2 |
| Hypokalemia | SUBJECTS | 1 ( 2.3%) |
| •• | | 1 |
| Mucositis | SUBJECTS | 2 ( 4.7%) |
| | EPISODES : | 2 |
| Nausea | SUBJECTS | 5 ( 11.6%) |
| | | 5 |
| Neutrophil count decreased | | 3 ( 7.0%) |
| • | | 4 |

Table 15.2. Adverse Events by Grade. Descriptive Statistics. Safety Analysis Set.

| Grade | | |
|-----------------------------------|----------|-------------|
| Term | | Total |
| D1-b-1-b dd | | |
| Platelet count decreased | | 2 ( 4.7%) |
| | EPISODES | |
| Serum Urea Increased | | 1 ( 2.3%) |
| Ti-i+i- | EPISODES | |
| Transaminitis | | 2 ( 4.7%) |
| W | EPISODES | |
| Vomiting | | 4 ( 9.3%) |
| | EPISODES | |
| White Blood Cells Decreased | | 1 ( 2.3%) |
| | EPISODES | 2 |
| Grade 2 | | - 4 |
| Anemia | | 5 ( 11.6%) |
| | EPISODES | |
| Asthenia | | 15 ( 34.9%) |
| | EPISODES | |
| Mucositis | | 2 ( 4.7%) |
| | EPISODES | |
| Nausea | | 3 ( 7.0%) |
| | EPISODES | |
| | | 7 ( 16.3%) |
| | EPISODES | |
| Palmar-Plantar Erythrodysesthesia | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | |
| Skin Disorders | | 2 ( 4.7%) |
| | EPISODES | |
| Urinary Tract Infection | | 3 ( 7.0%) |
| | EPISODES | |
| Vomiting | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | |
| White Blood Cells Decreased | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 2 |
| Grade 3 | | |
| Anemia | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Asthenia | SUBJECTS | 5 ( 11.6%) |
| | EPISODES | 5 |
| Mucositis | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 2 |
| Nausea | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |

Table 15.2. Adverse Events by Grade. Descriptive Statistics. Safety Analysis Set.

| Grade<br>Term | | Total |
|-----------------------------------|----------|------------|
| Neutrophil count decreased | SUBJECTS | 4 ( 9.3%) |
| | EPISODES | |
| Platelet count decreased | SUBJECTS | |
| | EPISODES | - |
| Respiratory Infection | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Transaminitis | SUBJECTS | 2 ( 4.7%) |
| | EPISODES | 2 |
| Vomiting | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Grade 4 | | |
| Neutrophil count decreased | SUBJECTS | 6 ( 14.0%) |
| | EPISODES | 6 |
| Unknown | | |
| Hypersensitization To Trabectidin | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Nausea | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |
| Neutrophil count decreased | SUBJECTS | 1 ( 2.3%) |
| - | EPISODES | |
| Platelet count decreased | SUBJECTS | 1 ( 2.3%) |
| | EPISODES | 1 |

Figure 3. Adverse Events by Grade. Descriptive Statistics. Safety Analysis Set.



-----

Table 15.6 Adverse Events by Highest grade per patient by Grade group. Descriptive Statistics. Safety Analysis Set.

| Haematology | | | | |
|---|---|---|---|---|
| Term | | I-II | | IV |
| Haematological | | | | |
| Neutrophil count decreased | 15 ( 34.9%) | 9 ( 20.9%) | 4 ( 9.3%) | 6 ( 14.0%) |
| Anemia | 10 ( 23.3%) | 9 ( 20.9%) | 1 ( 2.3%) | 0 |
| Platelet count decreased | 5 ( 11.6%) | 2 ( 4.7%) | 3 (7.0%) | 0 |
| White Blood Cells Decreased | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Non-Haematological | | | | |
| Asthenia | 21 ( 48.8%) | 19 ( 44.2%) | 5 ( 11.6%) | 0 |
| Nausea | 9 ( 20.9%) | 8 ( 18.6%) | 1 ( 2.3%) | 0 |
| Mucositis | 6 ( 14.0%) | 4 ( 9.3%) | 2 ( 4.7%) | 0 |
| Vomiting | 6 ( 14.0%) | 5 ( 11.6%) | 1 ( 2.3%) | 0 |
| Transaminitis | 4 ( 9.3%) | 2 ( 4.7%) | 2 ( 4.7%) | 0 |
| Urinary Tract Infection | 3 ( 7.0%) | 3 (7.0%) | 0 | 0 |
| Constipation | 2 ( 4.7%) | 2 ( 4.7%) | 0 | 0 |
| Hypertension | 2 ( 4.7%) | 2 ( 4.7%) | 0 | 0 |
| Skin Disorders | 2 ( 4.7%) | 2 ( 4.7%) | 0 | 0 |
| Abdominal pain | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Alopecia | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Dissociated Cholestasis | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Dysuria | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| General Muscular Pain | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Headache | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Hip or exia | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Hyp okalemia | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Palmar-Plantar Erythrodysesthesia | 1 ( 2.3%) | 1 ( 2.3%) | 0 | 0 |
| Respiratory Infection | 1 ( 2.3%) | 0 | 1 ( 2.3%) | 0 |

### 11. Discussion

### 11.1 Key results

- Between November 2021 and June 2022, 43 patients were recruited with median age 74 years (70-86).
- At initial diagnosis, most common FIGO stages were IIIC (51.2%), IVB (11.6%), and IIIB (7.0%).
- Before trabectedin+PLD (baseline):
- Patients had ECOG performance status 0, 1, or 2 (34.1%, 41.5%, and 9.8%) and 81.4% had measurable disease.
- The median number of previous lines was 2 (1-6).
- The initial dose of trabectedin was  $1.1 \text{ mg/m}^2$  in 76.7% of patients (16.3% with <1.1 and 4.7% with  $>1.1 \text{ mg/m}^2$ ) while 76.7% of patients had PLD at 30 mg (18.6% with <30 mg and 2.3% with >30 mg).
- The median of trabectedin+PLD cycles was 5 (1-21) and 53.5% of patients had at least one cycle delayed.
- All patients ended treatment for the following reasons: patient's decision (7.0%), doctor's decision (23.3%), disease progression (39.5%), toxicity (23.83%) and 7.0% due to other factors.
- Median PFS for the trabectedin+PLD combination was 7.7 months (95% CI 4.4-9.4) with best overall response rates of 4 CR (9.3%), 14 PR (32.6%), 13 SD (30.2%), and 5 PD (11.6%).
- Median overall survival (OS) was 19.5 months (95% CI 12.8-27.2).
- Overall, the most common G3-4 hematological events were neutropenia (23.3%), thrombocytopenia (7.0%), and anemia (2.3%), being asthenia (11.6%), mucositis (4.7%), and transaminitis (4.7%) the most frequent G3 non-hematological toxicities.

### 11.2 Limitations

Potential study limitations included:

- Heterogeneous population in terms of baseline characteristics (retrospective study)
- Limited follow-up and missing data

### 11.3 Interpretation

This study demonstrated that the safety profile of the trabectedin+PLD combination for elderly patients in real-life setting is manageable and efficacy results are comparable to those of previous clinical trials.

### 11.4 Generalisability

The safety and efficacy results of this study are comparable to those of previous clinical trials with trabectedin and PLD.

### 12. Other information

All patients participating in the study (accessible, alive patients who could be interviewed in the hospital) received a Patient Information Sheet (PIS) describing, in simple language, the goals, scope, procedures and relevant implications of the study.

The PIS integrated an Informed Consent Form (ICF) to be signed by the patient, which was indispensable for study participation (for accessible patients).

Written informed consent had to be given by each accessible/reachable patient before study initiation (prior to registration of the patient in the e-CRF). The PIS/ICF included the consent of patients for the collection and analysis of their clinical data.

Data of inaccessible/unreachable patients (dead, lost, etc.) could still be used according to the permissions of ethics committees and Spanish law, regarding the use of data in retrospective studies.

## 13. Conclusion

The safety profile of the trabectedin+PLD combination for elderly women in real-life setting is manageable and efficacy results are comparable to those of previous clinical trials. The results of this study are aligned with those reported in the literature for the general population.

### 14. References

- [1] De Angelis R, et al. EUROCARE-5 Working Group. Cancer survival in Europe 1999-2007 by country and age: results of EUROCARE--5-a population-based study. Lancet Oncol. 2014 Jan;15(1):23-34. doi: 10.1016/S1470-2045(13)70546-1.
- [2] Sabatier R, et al. Prognostic factors for ovarian epithelial cancer in the elderly: a case-control study. Int J Gynecol Cancer. 2015 Jun;25(5):815-22. doi: 10.1097
- [3] Von Gruenigen VE, et al. Chemotherapy completion in elderly women with ovarian, primary peritoneal or fallopian tube cancer An NRG oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2017;144(3):459-467. doi:10.1016/j.ygyno.2016.11.033
- [4] Falandri C, et al. EWOC-1: A randomized trial to evaluate the feasibility of three different first-line chemotherapy regimens for vulnerable elderly women with ovarian cancer (OC): A GCIG-ENGOT-GINECO study. J Clin Oncol 37, 2019, no. 15 suppl, 5508-5508.
- [5] Ovarian Cancer Incidence by International Agency for Research Cancer and WHO website: https://gco.iarc.fr/today/online-analysis-table?v=2018&mode=cancer&mode\_population=continents&population=900&populations=900&ke y=asr&sex=2&cancer=39&type=0&statistic=5&prevalence=0&population\_group=0&ages\_group% 5B%5D=0&ages\_group%5B%5D=17&group\_cancer=1&include\_nmsc=1&include\_nmsc\_other=1
- [6] Trabectedin (Yondelis®): Summary of Product Characteristics. http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_-\_Scientific\_Discussion/human/000773/WC500045836.pdf
- [7] Colombo N, et al. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent disease. Annals of Oncology. 2019. 30:672-705.
- [8] Pignata S, et al. A European, observational, prospective trial of trabectedin plus pegylated liposomal doxorubicin in patients with platinum-sensitive ovarian cancer. Oncologist. 2020 Dec 8. doi: 10.1002/onco.13630. Online ahead of print.
- [9] Monk BJ, et al. Trabectedin plus pegylated liposomal Doxorubicin in recurrent ovarian cancer. J Clin Oncol. 2010 Jul 1;28(19):3107-14. doi: 10.1200/JCO.2009.25.4037.
- [10] Oza AM, et al. Efficacy and Safety of Bevacizumab-Containing Therapy in Newly Diagnosed Ovarian Cancer: ROSiA Single-Arm Phase 3B Study. Int J Gynecol Cancer. 2017 Jan;27(1):50-58. doi: 10.1097
- [11] Sorio R, et al. Safety and efficacy of single-agent bevacizumab-containing therapy in elderly patients with platinum-resistant recurrent ovarian cancer: Subgroup analysis of the randomised phase III AURELIA trial. Gynecol Oncol. 2017;144(1):65-71. doi:10.1016
- [12] Dockery LE, et al. Tolerance and toxicity of the PARP inhibitor olaparib in older women with epithelial ovarian cancer. Gynecol Oncol. 2017;147(3):509-513. doi:10.1016

[13] Vergote I, et al. Safety analysis of trabectedin in combination with pegylated liposomal doxorubicin (PLD) vs PLD alone in ovarian cancer patients 65 years of age and older. vol 7 Supl (2) pages 458 (Abs. N° P8028) ECCO 15-34th ESMO European Society for Medical Oncology, september 20-24, 2009. Berlin. Eur J Cancer